**Clinical Study Protocol** Identification No.

EMR700568-012

**Title** 

Prospective observational long-term safety registry of Multiple Sclerosis patients who have participated in cladribine clinical

trials (PREMIERE)

**EudraCT Number** 

2009-017978-21

**Study Phase** 

Non-Experimental registry

**Investigational Medicinal** 

Cladribine Merck Europe 10 mg tablets

Product(s)

Cladribine is an adenosine deaminase-resistant analogue of deoxyadenosine that exerts its effect in MS via prolonged

suppression of peripheral lymphocyte counts

**Clinical Study Protocol** 

Version

20 July 2016 / Version 4.0 including amendment No.2

PPD

**Integrated Analysis Plan** 

Author

Coordinating Author

PPD Merck **Function Author** 

PP PPD

PPD

PPD

PPD

PPD

21 November 2018 / Version 1.0

**Integrated Analysis Plan** 

**Integrated Analysis Plan** 

**Date and Version** 

Reviewers

**Function** PPD Merck PPD Merck

Name PPD PPD

PPD

Merck PP

PPD PPD PPD

This document is the property of Merck KGaA, Darmstadt, Germany, or one of its affiliated companies. It is intended for restricted use only and may not - in full or part - be passed on, reproduced, published or used without express permission of Merck KGaA, Darmstadt, Germany or its affiliate.

Copyright © 2018 by Merck KGaA, Darmstadt, Germany or its affiliate. All rights reserved.

## **Approval Page**

**Integrated Analysis Plan:** EMR700568-012

Prospective observational long-term safety registry of Multiple Sclerosis patients who have participated in cladribine clinical trials (PREMIERE)

| Merck Responsible | Date | Signature |
|-------------------|--------------|--------------------|
| PPD | Via ELDORADO | O approval process |

| 1 | Table of Contents | |
|---|---|---|
| Integrated Analysi | is Plan | 1 |
| Approval Page | 2 | |
| 1 | Table of Contents | 3 |
| 2 | List of Abbreviations and Definition of Terms | 6 |
| 3 | Modification History | 7 |
| 4 | Purpose of the Integrated Analysis Plan | 8 |
| 5 | Objectives and Endpoints | 8 |
| 6 | Overview of Planned Analyses | 9 |
| 6.1 | Intermediate Analyses | 9 |
| 6.2 | Final Analysis | 9 |
| 7 | Changes to the Planned Analyses in the Clinical Study Protocol | 10 |
| 8 | Protocol Deviations and Analysis Populations | 12 |
| 8.1 | Definition of Protocol Deviations and Analysis Sets | 12 |
| 8.2 | Definition of Analysis Populations and Subgroups | 12 |
| 9 | General Specifications for Data Analyses | 13 |
| 9.1 | Treatment groups | 13 |
| 9.2 | Analysis Period | 14 |
| 9.3 | Identification of patients | 14 |
| 9.4 | Dictionary coding. | 14 |
| 9.5 | Study Day 1 | 15 |
| 9.6 | Registry Day 1 | 15 |
| 9.7 | Baseline | 15 |
| 9.8 | End of clinical trial | 15 |
| 9.9 | Last date in PREMIERE | 15 |
| 9.10 | Last ALC date with value in PREMIERE | 15 |
| 9.11 | Conversion factors | 15 |
| 9.12 | Handling of missing data | 16 |
| 9.13 | Presentation of continuous and qualitative variables | 16 |
| 9.14 | Significance level | 16 |
| 9.15 | Software(s) | 16 |
| 10 | Study Participants | 16 |

| Integrated Analysis Plan | |
|---|---|
| Disposition of Participants and Discontinuations | 16 |
| Protocol Deviations | 18 |
| Demographics and Other Baseline Characteristics | 18 |
| Demographics | 18 |
| Medical History | 19 |
| Previous Medications or Medications/Procedures in PREMIERE | 19 |
| Previous medications | 19 |
| Medications in PREMIERE | 19 |
| Disease Modifying Drugs in PREMIERE | 20 |
| Procedures in PREMIERE | 20 |
| Handling of Partial dates for Medications | 20 |
| Study intervention Compliance and Exposure | 21 |
| Efficacy Analyses | 21 |
| Safety Analyses | 21 |
| Primary Endpoints | 21 |
| Serious Adverse Events Related to Cladribine | 21 |
| Blood and Lymphatic System Disorders | 22 |
| Neoplasms Benign, Malignant, and Unspecified | 23 |
| Lymphopenia | 23 |
| Secondary Endpoints: Pregnancy | 26 |
| Adverse Events | 27 |
| All Adverse Events | 27 |
| Serious Adverse Events | 27 |
| Deaths, Other Serious Adverse Events, and Other Significant Adverse Events | 28 |
| Deaths | 28 |
| Adverse Event of Special Interest | 28 |
| AESI= Infections | 28 |
| AESI = Malignancies | 30 |
| Handling of Missing or Partial AE Dates (onset, resolution date) | 30 |
| Clinical Laboratory Evaluation | 30 |
| Vital Signs | 30 |
| Other Safety or Tolerability Evaluations | 30 |
| | Disposition of Participants and Discontinuations Protocol Deviations Demographics and Other Baseline Characteristics Demographics Medical History. Previous Medications or Medications/Procedures in PREMIERE Previous medications Medications in PREMIERE Disease Modifying Drugs in PREMIERE. Procedures in PREMIERE Handling of Partial dates for Medications Study intervention Compliance and Exposure Efficacy Analyses Safety Analyses Primary Endpoints Serious Adverse Events Related to Cladribine Blood and Lymphatic System Disorders Neoplasms Benign, Malignant, and Unspecified Lymphopenia Secondary Endpoints: Pregnancy Adverse Events All Adverse Events Serious Adverse Events Serious Adverse Events |

| Cladribine<br>EMR700568-012 | Integrated Analysis Plan |
|---|---|
| 16 | Analyses of Other Endpoints |
| 17 | References 31 |
| 18 | Appendices 32 |
| 18.1 | Pregnancy and neonatal topics (SMQ 20000185)32 |
| 18.2 | Adverse Events Related to Pregnancy |
| 18.3 | AESI: Opportunistic Infections 1 |
| 18.4 | AESI Herpes Zoster |
| 18.5 | Malignant or Unspecified Tumours (SMQ 20000091)4 |
| 18.6 | AESI: Malignancies |
| Table 1 | Changes from the planned analyses in the clinical study protocol 10 |
| Table 2 | Table header example |
| Table 3 | Identification 14 |
| Table 4 | Time intervals |
| Table 5 | List of MS-DMD. 20 |
| Table 6 | NCI-CTCAE Lymphopenia Grade |
| Table 7 | Time window for lymphocyte from first cladribine/placebo dose 24 |
| Table 8 | Time window for lymphocyte from the end of clinical trial25 |
| Table of Content | ts of Figure |
| Figure 1 | PREMIERE Registry Overview Diagram |

#### 2 List of Abbreviations and Definition of Terms

AE Adverse Event

ADR Adverse Drug Reaction

ATC Anatomical Therapeutic Chemical classification
CDISC Clinical Data Interchange Standards Consortium

CI Confidence Interval

CMQ Custom MedDRA query

(e)CRF (electronic) Case Report Form

CSR Clinical Study Report

CTCAE Common Terminology Criteria for Adverse Events

EMA European Medicines Agency

EudraCT European Union Drug Regulating Authorities Clinical Trials

FDA Food and Drug Administration

GCP Good Clinical Practice
GDS Global Drug Safety

GPP Good Pharmacoepidemiology Practices

HLGT High Level Group Term

HLT High Level Term

IAP Integrated Analysis Plan

ICH International Conference on Harmonization

IEC Independent Ethics CommitteeIRB Independent Review BoardISS Integrated Summary of Safety

KM Kaplan-Meier

LLN Lower limit of normal

MedDRA Medical Dictionary for Regulatory Activities

NA Not Applicable

NCI-CTCAE National Cancer Institute – Common Terminology Criteria for Adverse

Events

P1 Original cladribine clinical trial physician

P2 Usual health care provider
PRP Principal registry physician

## **Integrated Analysis Plan**

PT Preferred Term

RRMS Relapsing-remitting MS

SADR Serious Adverse Drug Reaction

SAE Serious Adverse Event SAP Statistical Analysis Plan

SDTM Study Data Tabulation Model SMQ Standard MedDRA query

SOC System Organ Class

SUSAR Suspected Unexpected Serious Adverse Reaction

TEAE Treatment-Emergent Adverse Event

TLF Tables, Listings, and Figures

WHO-DD World Health Organization Drug Dictionary

## **3** Modification History

| Unique<br>Identifier for<br>Version | Date of<br>IAP Version | Author | Changes from the Previous Version |
|---|---|---|---|
| NA | | | |

## 4 Purpose of the Integrated Analysis Plan

The purpose of this IAP (integrated analysis plan) is to document technical and detailed statistical specifications for the final analysis of data collected for protocol EMR700568-012 called PREMIERE. Results of the analyses described in this IAP will be included in the Clinical Study Report (CSR). Additionally, the planned analyses identified in this IAP will be included in regulatory submissions or future manuscripts. Any post-hoc, or unplanned analyses performed to provide results for inclusion in the CSR but not identified in this prospective IAP will be clearly identified in the CSR.

The IAP is based upon section 9 (Data Analysis and Statistics) of the study protocol and protocol amendments and is prepared in compliance with International Conference on Harmonization (ICH) E9 and Guidelines for Good Pharmacoepidemiology Practices (GPP). It describes analyses planned in the protocol and protocol amendments.

## 5 Objectives and Endpoints

| | | | ı |
|---|---|---|---|
| Objectives | Endpoints (Outcome<br>Measures) | Endpoints (Outcome<br>Measures) Timeframe | IAP section |
| Primary | | | |
| To quantify and characterize the risk (cumulative incidence) of serious adverse drug reaction (SADR), including malignancies and serious infections To assess time to resolution of lymphopenia among registry participants with persistent lymphopenia To quantify and characterize the risk (cumulative incidence) of AE in the 'Blood and Lymphatic System Disorders' and 'Neoplasms Benign, Malignant, and Unspecified' System Organ Classes (SOCs) | Cumulative incidence of SADR, including malignancies and serious infections Time to resolution of lymphopenia, among registry participants with persistent lymphopenia Cumulative incidence of all AEs in the "Blood and Lymphatic System Disorders" System Organ Class (SOC) and in the "Neoplasms Benign, Malignant, and Unspecified" SOC | AE crude incidence from Registry Day 1 to End of registry Time to resolution of lymphopenia, for participants with ongoing lymphopenia at the end of clinical trial AE crude incidence from Registry Day 1 to End of registry | • Section<br>15.1.1<br>• Section<br>15.1.4<br>• Section<br>15.1.2 &<br>15.1.3 |
| Secondary | | | |
| To assess pregnancy outcomes, including congenital malformations or other important health conditions in the offspring born to women exposed to oral cladribine Pregnancy outcomes, including congenital malformations, spontaneous abortion, elective abortion, stillbirth, ectopic pregnancy, molar pregnancy, and other important health conditions in the offspring | | Number of patients with<br>pregnancies from Registry<br>Day 1 to End of registry and<br>descriptive statistics of<br>pregnancy outcomes | • Section 15.2 |

## **6** Overview of Planned Analyses

## **Summary of PREMIERE registry**

The PREMIERE study is an ongoing prospective observational long-term safety registry of patients who have participated in at least one of the 5 cladribine clinical trials (namely CLARITY [25643], CLARITY EXT [27820], ONWARD [26593], ORACLE [28821] and the pantoprazole drug-drug interaction [DDI] phase I study [27967]. These 5 studies are referred throughout this document under the general term "clinical trials".

The original objectives of the PREMIERE registry were to monitor long-term safety events in a clinical trial population to produce long-term safety data in order to better characterize the potential safety risks of oral cladribine, and to build an evidence-based risk minimization strategy. The study was amended with simplification and including restriction to serious adverse drug reactions (SADR), selected AEs (all AEs in the 'Blood and Lymphatic System Disorders' and 'Neoplasms Benign, Malignant, and Unspecified' SOCs) and reduction of frequency of assessments. The duration of follow-up in the registry is up to the end of the registry or 8 years after the subject's first enrolment into a cladribine clinical trial, whichever occurs first. Last patient last visit for the final analysis was on October 25<sup>th</sup>, 2018.



Figure 1 PREMIERE Registry Overview Diagram

#### 6.1 Intermediate Analyses

Two intermediate safety synoptic reports have been performed while the study was ongoing (REF. CSR items #1 and #2). The data cut-off for the first analysis was 20 February 2015 and the cut-off for the second analysis was 15 May 2017.

## **6.2** Final Analysis

All final, planned analyses identified in the Clinical Study Protocol and in this IAP will be performed only after the last participant has completed the study (following protocol definition) with all study data in-house, all data queries resolved as much as possible, and the database locked.

# 7 Changes to the Planned Analyses in the Clinical Study Protocol

As usual, Statistical Analysis Plans are more detailed than relevant sections of the Study Protocols; such additions and refinements are therefore not mentioned in this section. Instead, only true deviations from statements in the study protocol are listed together with a brief rationale.

Table 1 Changes from the planned analyses in the clinical study protocol

| Protocol Section: Item | Protocol definition | Changes implemented in the SAP |
|---|---|---|
| Section 5.6: Study Cohort | There will be no control/comparison group | "Never exposed to Cladribine" group will be considered as reference for a long-term non-treated population. |
| Section 9.2.2:<br>Treatment/Analysis periods | The most relevant analysis period will be the cumulative analysis period, which starts from the date of first dose of clinical trial medication to the end of the registry follow-up. In addition of the cumulative period, three treatment periods are identified: a) the initial treatment period, from the date of first dose of clinical trial medication to end of the clinical trial participation; b) the extension treatment period (when subjects elects to enroll in a cladribine extension trial) from the date of first dose of cladribine to the end of extension trial participation, c) and the registry study period (where subjects do not receive any experimentally assigned treatment) from the date of enrollment into the registry to the end of registry participation. The primary analysis will correspond to the cumulative analysis period, which starts from the date of first dose of clinical trial medication to the end of registry follow-up. | The primary analysis will <b>NOT</b> start from the date of first dose of clinical trial medication to the end of registry follow-up. Reporting for the clinical trial period has been presented in each individual study CSR. In the Integrated Summary of Safety (ISS) for the proposed indication of Cladribine in the treatment of adult patients with relapsing forms of Multiple Sclerosis (RMS), long-term data available at the cut-off date of 15 May 2017 has already been presented exhaustively, including all subjects – those enrolled and those not enrolled in Premiere. In order to focus on the long-term safety events that were collected during the registry follow-up, the analysis period for the safety analysis population will be the time from the end of clinical trial + 1 day to the last date in PREMIERE registry. In addition, two analysis periods for the lymphocyte analysis population will be defined: • The time from first dose of cladribine/placebo* in clinical trials to the last Absolute Lymphocyte Count (ALC) date with a value available in PREMIERE registry |

| | | The time from first ALC date with value in PREMIERE registry to the last ALC date with a value available in PREMIERE registry * A subject who switches treatment from placebo to cladribine in subsequent studies/periods will be considered from first dose of cladribine and the placebo period will not be considered. |
|---|---|---|
| Section 9.2.2<br>Treatment/Analysis periods | Demographic characteristics (e.g., age, sex) at baseline of the registry will be described using descriptive statistics for continuous variables or proportions for categorical variables at entry into the registry. Summaries will be provided by region/country. | Demographic characteristics will not be summarized by region/country. Instead, based on the understanding of the protocol, summary statistics for the number of subjects by country will be provided. |
| Section 9.2.1 General<br>Considerations | Time to resolution of persistent lymphopenia will be estimated using the life table methodology. | The time to resolution of lymphopenia (duration of lymphopenia episode) has already been presented in the ISS using the product-limit method of Kaplan and Meier. This analysis will not be repeated. The time to resolution of lymphopenia for participants with ongoing lymphopenia at end of clinical trial will be analyzed using descriptive statistics. |
| Section 9.2.1 General<br>Considerations | The main analysis will be to estimate cumulative incidence rates using life-table methodology. | The main analysis of adverse events will be done on the period from the end of clinical trial + 1 day to the last date in PREMIERE registry. The life-table methodology will not be used. Rather, the crude incidence will be presented with the corresponding 95% confidence interval. The time to first event from the first dose of cladribine has already been presented in the ISS following the Kaplan-Meier methodology for AESI infections and malignancies. Therefore, it will not be repeated here. |

| Section 10.2 Subject information and informed consent | Subjects who refuse to enroll in the registry will be asked to sign consent (see CRF: Data Release Participant only) for use of their clinical trial data to compare registry non-participants with registry participants in terms of demographics, cancer risk factors and severity of MS. | Comparison of registry participant's vs non-registry participants will not be performed due to very strong sample size imbalance between the 2 groups. Indeed as the registry target population was of 2175 subjects, 1161 patients enrolled as full participants and 22 refused and signed the data release consent form only. |
|---|---|---|
|---|---|---|

### **8** Protocol Deviations and Analysis Populations

## 8.1 Definition of Protocol Deviations and Analysis Sets

Important protocol deviations are protocol deviations that might significantly affect the completeness, accuracy, and/or reliability of the study data or that might significantly affect a participant's rights, safety, or well-being.

For this study, important protocol deviations will be identified and confirmed at the protocol deviation review meetings.

## 8.2 Definition of Analysis Populations and Subgroups

The registry target population includes all subjects who participated in Sponsor oral cladribine Phase I to III clinical trials in MS associated with a protocol approved prior to the time of submission of the marketing application and completed (last patient, last visit) after November 2008. This corresponds to five clinical trials (protocol number/study name):

- 25643/CLARITY
- 26593/ONWARD
- 27820/CLARITY EXTENSION
- 27967/Pantoprazole DDI
- 28821/ORACLE MS

Subjects will be analyzed according to their actual exposure to oral cladribine. There will be no per-protocol analysis population excluding patients with protocol deviations.

#### **Safety Analysis Population (SAF)**

The Safety Analysis Population will consist of all subjects from studies CLARITY, CLARITY EXT, ORACLE MS and ONWARD who are enrolled in the PREMIERE registry as full participants.

## **Lymphocyte Analysis Population**

The lymphocyte analysis population consists of all subjects from SAF with at least one absolute lymphocyte count (ALC) value in PREMIERE, with an associated ALC date after the end of clinical trial.

#### **DDI Safety Set**

The **DDI** Safety Set will include all subjects from the Pantoprazole DDI study who are enrolled in the PREMIERE registry as full participants. In this study, subjects received two single doses of 10 mg cladribine separated by a wash-out of at least 10 days and two 40 mg doses of pantoprazole on two consecutive days. Data from the DDI Safety Set will be presented in listings only.

## 9 General Specifications for Data Analyses

## 9.1 Treatment groups

Analyses will be performed on the "as treated principle", where patients are allocated to the treatment group that they actually received in the clinical trial studies (which may be different from the study treatment to which they were randomized to).

Patients are assigned to the following treatment groups according to their actual treatment in one of the studies CLARITY alone, ONWARD, CLARITY/CLARITY EXTENSION, ORACLE MS, Pantoprazole DDI.

- Never exposed to cladribine: if a subject has taken only placebo (or placebo +IFN-β) in studies, then her/his data becomes part of the "Never exposed to cladribine" treatment group. A subject who switches treatment from placebo to cladribine in subsequent studies/periods will not be considered in this group.
- **Exposed to cladribine**: patients with at least one dose of cladribine. Subjects who were on placebo during the clinical trial and switched to cladribine in the extension study will contribute to the treatment group "Exposed to cladribine" from the moment they initiate cladribine.

An example of the header for table outputs is presented below.

Table 2 Table header example

| | Never exposed to<br>Cladribine<br>(N=XXXX) | Exposed to Cladribine (N=XXXX) | Total<br>(N=XXXX) |
|---|---|---|---|
| Safety Analysis<br>Population | xxx (100.0) | xxx (100.0) | xxx (100.0) |

## 9.2 Analysis Period

#### Analysis period for Safety Analysis Population and the DDI Safety Set

The analysis period for SAF and the DDI Safety Set is the time from the end of clinical trial + 1 day to the last date in PREMIERE.

#### Analysis period for Lymphocyte Analysis Population

Two analysis periods for lymphocyte analysis population are defined:

- 1. The time from first dose of cladribine/placebo\* in clinical trials to the last absolute lymphocyte count (ALC) date with a value available in PREMIERE registry.
- 2. The time from first ALC date with a value in PREMIERE registry to the last ALC date with a value available in PREMIERE registry.
- \* A subject who switches treatment from placebo to cladribine in subsequent studies/periods will be considered from first dose of cladribine and the placebo period will not be considered.

## 9.3 Identification of patients

Patients are identified by their unique subject number taken from the subject ID in their first study. Other variables are created to distinguish their previous trial origin.

Table 3 Identification

| Unique Subject Identifier<br>(USUBJID) | First Previous<br>Study Identifier | Last Previous<br>Study Identifier<br>(if diff) | Previous Clinical Trial |
|---|---|---|---|
| PPD | PPD | | CLARITY only |
| PPD | PPD | | ONWARD |
| PPD | PPD | PPD | CLARITY/CLARITY EXTENSION |
| PPD | PPD | | Pantoprazole DDI |
| PPD | PPD | | ORACLE MS |

#### 9.4 Dictionary coding

The Adverse events (AEs) and Medical History will be coded to MedDRA version 21.0. Concomitant medications will be upgraded with WHO Drug Dictionary version March 2018 (WHODRUG B2 MARCH2018).

## 9.5 Study Day 1

Study Day 1 is the day of start of first study drug intervention (placebo or cladribine). For patients in the sequence placebo-cladribine, the placebo period is ignored and Study Day 1 is at the start of cladribine. The day before is Study Day -1 (no Study Day 0 is defined).

## 9.6 Registry Day 1

Registry Day 1 is defined as the end of clinical trial +1 day. The day before is Registry Day -1 (no Registry Day 0 is defined).

#### 9.7 Baseline

Baseline is defined as registry baseline, which is the last assessment prior to or at Registry Day 1.

Unless specified, the demographics at baseline will be computed considering the last assessment prior to or at Registry Day 1.

#### 9.8 End of clinical trial

The end of the clinical trial is defined as the last date of data collection from the last cladribine clinical trials.

#### 9.9 Last date in PREMIERE

Last date in PREMIERE is the last date from any datasets including death and AE start date.

Programming rule to cover possible unclean data:

For subjects who died, last date in PREMIERE is the date of death and all data collected after date of death are ignored.

## 9.10 Last ALC date with value in PREMIERE

Last ALC date with an associated value (value not missing) in the PREMIERE registry is considered.

Programming rule to cover possible unclean data:

The last ALC date with value in PREMIERE is defined as the last ALC date with value after the end of clinical trial.

#### 9.11 Conversion factors

Unless specified, the following conversion factors will be used to convert days into months or vears:

• 1 year = 12 months = 365.25 days

## 9.12 Handling of missing data

Several attempts are to be made to contact subjects and to limit missing data (see protocol section 9.3.1). There will be no imputation for missing data.

#### 9.13 Presentation of continuous and qualitative variables

#### **Continuous and qualitative variables:**

Continuous variables will be summarized using descriptive statistics, i.e.

- number of subjects (N),
- number of subjects with non-missing values,
- mean, standard deviation,
- median, 25th Percentile 75th Percentile (Q1-Q3),
- minimum, and maximum.

#### Qualitative variables:

Qualitative variables will be summarized by counts and percentages. Unless otherwise stated, the calculation of proportions will be based on the number of subjects in the analysis set of interest. Therefore, counts of missing observations will be included in the denominator and presented as a separate category.

## 9.14 Significance level

There are no plans for any statistical inference. This study will adhere to the Guidelines for Good Pharmacoepidemiology Practices (GPP). Accordingly, data evaluations and interpretations will be based on point estimates and 95% confidence intervals (CI) for the evaluation of the statistical precision around the point estimate.

#### 9.15 Software(s)

Analyses will be performed using SAS® Software version 9.4 or higher.

#### 10 Study Participants

The subsections in this section describe the specifications for reporting participant disposition and study discontinuations.

#### 10.1 Disposition of Participants and Discontinuations

Number of subjects screened (full participant + data release participant), number of subject enrolled (full participant), number of subjects in the SAF and in the DDI Safety Set will be presented by treatment group (never exposed to cladribine and exposed to cladribine) and total.

The number of subjects in the Lymphocyte Analysis Population will be summarized based on the SAF.

Study status will be summarized on the SAF by treatment group and total, presented as

- Completed or
- Discontinued.

Reason for study discontinuation will be summarized. Percentages will be presented with respect to the number of full participants.

## Programming rule

Programming rule to cover potential unclean data: Patients who died will be set to study status "Discontinued", with reason ="Death".

Time since end of clinical trial, time since first dose will be summarized in weeks as a continuous variable and in cumulative intervals and in time intervals with the following categories:

Table 4 Time intervals

| Cumulative intervals | Time intervals |
|------------------------|----------------------------------|
| Less than 12 weeks | 1 to 84 days (12 weeks) |
| At least 12 weeks | 85 to 168 days (24 weeks) |
| At least 24 weeks | 169 to 252 days (36 weeks) |
| At least 36 weeks | |
| | 253 to 336 days (48 weeks, 1y) |
| At least 48 weeks, 1y | 337 to 420 days (60 weeks) |
| At least 60 weeks | 421 to 504 days (72 weeks) |
| At least 72 weeks | 505 to 588 days (84 weeks) |
| At least 84 weeks, 2y, | 589 to 672 days (96 weeks, 2y) |
| At least 96 weeks, 3y, | 673 to 1008 days (144 weeks, 3y) |
| Etc. | Etc. |

Patient-year will be computed as the sum per group of the time since end of the clinical trial, in years. Patient-year will be presented per treatment group and total.

Reporting on study status will be done for SAF.

The disposition table will be repeated by

- CLARITY only
- CLARITY/CLARITY EXTENSION
- ORACLE MS
- ONWARD

#### 10.2 Protocol Deviations

Important protocol deviations will be summarized by type of deviation. In addition, a listing of PREMIERE important protocol deviations will be provided.

#### **Programming Note**

Information will be taken from SDTM.DV dataset.

## 11 Demographics and Other Baseline Characteristics

Summaries will be presented on SAF by treatment group and total.

## 11.1 Demographics

The following variables will be presented. Variables with \* are computed prior to first clinical trial study.

- Age at baseline (Registry Day 1), years and in categories (<= 40 y, >40 y)
- Sex (male, female)\*
- Race\*
- Region: America US, America non-US\*\*, Western Europe, Australia, Eastern Europe, Russia, ROW\*
  - \*\*America non-US includes Canada and all countries from South America.
- Previous clinical trial: CLARITY only, ONWARD, CLARITY/CLARITY EXTENSION, ORACLE MS.
- Time since last Cladribine/Placebo dose (weeks)
- Total cumulative dose (mg/kg): summary statistics and in categories 0, >0-3.5, >3.5-5.25, >5.25-7.0, >7.0-8.75, >8.75.

## 11.2 Medical History

No reporting will be done.

## Previous Medications or Medications/Procedures in PREMIERE

Medications in PREMIERE will be presented by Category, Therapeutic group (ATC level 2) and Preferred Name, per treatment group and total, using crude incidence:

Crude incidence, in % = (number of subjects with at least one medication / total number of subjects) \*100.

The following categories as reported in the CRF will be presented:

- MS-Related Immunomodulators and Immunosuppressants programming note CM.CMSPID = 101-199
- MS-Related Symptomatic Medications, including pain control programming note CM.CMSPID = 201-299
- MS-Related Antidepressants programming note CM.CMSPID = 301-399
- OTHER MS- AND NON-MS-RELATED programming note CM.CMSPID = 401-499

#### 12.1 Previous medications

Reporting of previous medications was done previously in each initial study CSR. No reporting will be done for the PREMIERE CSR.

#### 12.2 Medications in PREMIERE

Reporting will be done for SAF.

**Medications in PREMIERE** are medications (other than cladribine or placebo medications) which are taken by subjects at any time after (>) the end of clinical trial.

Data collection will be derived from PREMIERE dataset Concomitant Medication panel (SDTM.CM). Specifically, medications used during pregnancy collected for female partner of male patients will not be included (SDTM.CM CMCAT = "over the counter medications", "prescription medications").

## 12.2.1 Disease Modifying Drugs in PREMIERE

MS-disease modifying drugs (DMDs) drugs are defined by **custom selection** based on all concomitant medication collected.

Table 5 List of MS-DMD

| Preferred Term (WHODD) |
|----------------------------|
| ALEMTUZUMAB |
| BETASERON /01229701/ |
| DIMETHYL FUMARATE |
| FINGOLIMOD |
| FINGOLIMOD HYDROCHLORIDE |
| FUMARIC ACID |
| GLATIRAMER ACETATE |
| INTERFERON BETA |
| INTERFERON BETA-1A |
| INTERFERON BETA-1B |
| MITOXANTRONE |
| MITOXANTRONE HYDROCHLORIDE |
| NATALIZUMAB |
| PEGINTERFERON BETA-1A |
| RITUXIMAB |
| TERIFLUNOMIDE |

Note: the final list of medications may be revised after database lock. Any changes from the list above will be described in the CSR.

#### 12.3 Procedures in PREMIERE

Procedures are not coded in PREMIERE. No reporting will be done.

## **12.4** Handling of Partial dates for Medications

Missing and partial dates will be imputed considering the fact that medication may be considered as medication taken concomitantly to PREMIERE registry.

- Start missing day will be imputed to be 1 and start missing month will be imputed to be January.
- End missing day will be imputed to be the last day of the month. End missing month will be imputed to the last month of the year. In case of death, imputation rules will assure that no end dates are imputed after death.
- No imputation for complete start date and end date missing (day, month and year), and therefore medication will be ignored.

- If start date is completely missing (i.e. day, month, year missing) and end date is known or partially known then the start date will be imputed to be the Registry Day 1 minus one day if prior to end date, otherwise equal to end date.
- Complete end date missing (day, month and year) and partial or complete start date then will be imputed to be the last study assessment date.

## 13 Study intervention Compliance and Exposure

Not Applicable (please see section 7).

14 Efficacy Analyses

Not Applicable.

15 Safety Analyses

15.1 Primary Endpoints

#### 15.1.1 Serious Adverse Events Related to Cladribine

Reporting will be done for SAF.

The objective is "to quantify and characterize the risk (cumulative incidence) of SADR, including malignancies and serious infections".

#### Definition

The primary endpoint will be selected considering any serious adverse event characterized as Probable or Possible in the relationship to cladribine. Malignancies and serious infections will be considered in this endpoint only if the characteristics "serious" and "related" ("probable" or "possible") are applicable.

Following protocol section 8.5.1.2, "an adverse drug reaction (ADR) is a response to a medicinal product which is noxious and unintended, and which occurs at doses normally used in man for prophylaxis, diagnosis, or therapy of disease or for the restoration, correction, or modification or physiological functions. Response in this context means that a causal relationship between a medicinal product and an adverse event is at least a reasonable possibility".

The treating physician or other relevant concerned health care provider are asked to assess the relationship of the AEs to cladribine using the following definition, similar in all studies:

• Probable: A causal relationship is clinically/biologically highly plausible, and there is a correlation between the onset of the SAE and administration of cladribine, and between withdrawal of cladribine and resolution of the SAE.

- Possible: A causal relationship is clinically/biologically plausible and there is a correlation between the onset of the SAE and administration of cladribine.
- Unlikely: A causal relationship is improbable, and another documented cause of the SAE is most plausible.
- Unrelated: A causal relationship can be definitively excluded, and another documented cause of the SAE is most plausible.

The following statistics will be presented:

- Patient-year is the sum of the time since the end of clinical trial, expressed in years. Display with 1 decimal.
- m is the number of unique events. A unique event is a unique Preferred Term and date of onset per subject.
- n is the number of subjects with at least one event
- N is the total number of subjects in the treatment group
- AE (%) is the crude incidence. Display with 1 decimal.
  - o AE(%) = (number of subjects with at least one event / total number of subjects) \*100
- 95% Confidence Interval (CI) for the crude incidence within group for patients with at least one AE. The 95% Confidence Interval of the AE will be computed using the exact Clopper-Pearson confidence interval formula for binomial proportions (REF. Clopper item #3).

#### **Statistics description**

The following statistics per treatment group and total will be presented:

- Summary: Patient-years will be provided in the summary table. In addition, number of unique event, number of patients with at least one AE, crude incidence (%), 95% CI of the crude incidence. All these statistics will be repeated for AE leading to death and serious AE.
  - Note: SADR is a serious AE by definition. Therefore, only SADR and SADR leading to death will be presented.
- By SOC/ HLGT/ HLT/PT: Number of patients with the AE and crude incidence (%) will be presented by system organ class (SOC), High Level Group Term (HLGT), High Level Term (HLT), and preferred term (PT).

## 15.1.2 Blood and Lymphatic System Disorders

Reporting will be done for SAF.

Any adverse event preferred term belonging to the MedDRA SOC="Blood and Lymphatic System Disorders" will be selected.

Statistics as presented for section 15.1.1, Serious Adverse Events Related to Cladribine, will be repeated.

## 15.1.3 Neoplasms Benign, Malignant, and Unspecified

Reporting will be done for SAF.

Any adverse event preferred term belonging to the MedDRA SOC="Neoplasms Benign, Malignant, and Unspecified" will be selected.

Analyses as presented for SOC="Blood and Lymphatic System Disorders" will be repeated.

## 15.1.4 Lymphopenia

Unless specified, reporting will be done for the Lymphocyte Analysis Population.

Evolution of absolute lymphocyte count (ALC) and specifically lymphopenia is of primary interest for treatment with cladribine.

ALC will be tabulated by grade using the NCI-CTCAE version v3.0, and lymphopenia grades are defined as follows:

Table 6 NCI-CTCAE Lymphopenia Grade

| Laboratory<br>Toxicity | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| ALC Decreased | <lln 800="" mm<sup="" –="">3</lln> | <800 – 500/mm³ | <500 - 200/mm <sup>3</sup> | <200/mm <sup>3</sup> |
| | <lln 0.8="" x<br="" –="">10<sup>9</sup>/L</lln> | <0.8 – 0.5 x 10 <sup>9</sup> /L | <0.5 – 0.2 x 10 <sup>9</sup> /L | < 0.2 x 10 <sup>9</sup> /L |

#### Change from first cladribine/placebo dose

Data collected from first cladribine/placebo dose [Study Day 1] to the last ALC value in PREMIERE will be presented and summarized on a continuous manner (change from Study Day 1 and absolute value) and by grade, over time.

ALC Study Baseline is defined by the latest ALC value prior or equal to first cladribine/placebo dose [Study Day 1].

Over-time target point will be presented using visit window computed relative to Study Day 1, as presented below.

In case multiple samples are collected in the same window, the value closest to the target day will be used for analysis, where the target day is the middle of the time window. If there are two values with the same time before and after the target day, the earlier (first) value will be used for analysis.

Table 7 Time window for lymphocyte from first cladribine/placebo dose

| Evaluation | Target point (day) | Interval for analysis (Day) |
|---|---|---|
| ALC Study Baseline | Study Day 1 | Last value prior to or equal to Study Day 1 |
| Week 2 | 14 | [2;23] |
| Week 5 | 35 | [24 ; 47 ] |
| Week 9 | 63 | [48; 77] |
| Week 13 | 91 | [78; 103] |
| Week 16 | 112 | [104 ; 130 ] |
| Week 24 | 168 | [131 ; 203 ] |
| Week 36 | 252 | [204 ; 287 ] |
| Week 44 | 308 | [288 ; 329 ] |
| Week 48 | 336 | [330 ; 350 ] |
| Week 52 | 364 | [351 ; 376 ] |
| Week 55 | 385 | [377 ; 399 ] |
| Week 60 | 420 | [400 ; 461 ] |
| Week 72 | 504 | [462 ; 546 ] |
| Week 84 | 588 | [547 ; 630 ] |
| Week 96 | 672 | [631; 686] |
| Week 101 | 707 | [687 ; 721] |
| Week 105 | 735 | [722 ; 784] |
| Week 120 | 840 | [785 ; 924 ] |
| Week 144 | 1008 | [925 ; 1092 ] |
| Week 168 | 1176 | [1093 ; 1260 ] |
| Week 192 | 1344 | [1261 ; 1428 ] |
| Week 216 | 1512 | [1429 ; 1596 ] |
| And every 24 weeks If | | |
| needed | | |

#### Change from the end of clinical trial

A summary table of ALC similar to change from first cladribine/placebo dose will be presented.

Data collected from last value from the end of clinical trial to the last ALC value in PREMIERE will be presented and summarized on a continuous manner (absolute value only) and by grade, over time.

ALC Registry Baseline is defined as the first ALC date with a value on or after the end of clinical trial +1 day [Registry Day 1].

Programming rule to cover possible unclean data:

If first ALC date in PREMIERE is before the end of clinical trial, ALC Registry Baseline is defined as the first ALC value in PREMIERE on or after the end of clinical trial + 1 day.

A new set of time window are presented below using visit window computed relative to ALC Registry Baseline.

If more than 1 value is available for a particular time window for the same subject, the first value in the time window will be considered.

Table 8 Time window for lymphocyte from the end of clinical trial

| Evaluation | Interval for analysis (day) |
|---|---|
| Last value from last clinical trial | |
| ALC Registry Baseline | First ALC date with value in PREMIERE registry |
| Week 12 | [2 - 98] |
| Week 24 | [99 - 182] |
| Week 36 | [183 - 266] |
| Week 48, 1y | [267 - 350] |
| Week 60 | [351 - 434] |
| Week 72 | [435 - 518] |
| Week 84 | [519 - 602] |
| Week 96, y2 | [603 - 700] |
| Week 144, y3 | [701 – 1036] |
| Etc. | [1037 – weekN*7+4*7] |

#### Lymphopenia grade and MS-DMD

Best and Worst ALC grades will be presented in relation to use of MS-DMD medication. For subjects with MS-DMD medications reported at least once after end of clinical trial, the best and worst ALC grade will be selected on or after (>=) the first MS-DMD.

The Worst and the Best grade will be summarized overall and by treatment group. Subjects who are not taking MS-DMD from the end of clinical trial +1 day to the end of PREMIERE will be excluded from the analysis.

#### Resolution of lymphopenia computed with observed ALC value

Subjects who complete or drop out at the end of the clinical trial with an unresolved lymphopenia will be presented, together with their outcome in PREMIERE registry. The outcome can be resolved or unresolved.

An unresolved lymphopenia is defined for a subject who left the end of a clinical trial without returning to normal or grade 1 ALC value after an episode of grade 3 or 4 lymphopenia. A grade 3 or 4 lymphopenia episode is defined by a start/end date. Start= ALC>=grade 3, post baseline, End = following normal (grade 0) or grade 1.

The duration (in months) of the resolved episodes (out of the unresolved at end of clinical trial period) will be summarized. In addition, use of MS-DMDs prior to resolution will be presented.

## Resolution of lymphopenia computed using CRF tick box

Reporting will be done for SAF. This is an exception, to include the largest possible information available.

The number of subjects with declared Grade 3 or 4 lymphopenia at end of clinical trial [CRF Tick box], will be summarized together with their outcome in PREMIERE. The outcome in PREMIERE will be computed from those with at least one grade 0/1 in PREMIERE or with a CRF "resolution date".

Presentation per treatment group and total will be done.

#### Resolution of lymphopenia based on observed ALC value versus CRF tick box

A 2-by-2 table of number of subjects with and without resolution of lymphopenia at the end of clinical trial based on ALC value versus CRF Tick box will be presented.

In addition, a listing will be generated for subjects with unresolved lymphopenia at the end of clinical trial according to ALC grade, but with the CRF Tick box = "Resolved". The following variables will be displayed: Subject ID, cumulative dose of cladribine, previous clinical trial, treatment group (see section 9.1), all ALC values in PREMIERE with grade and date and tick box for resolved with date of resolved if available.

## 15.2 Secondary Endpoints: Pregnancy

Reporting will be done for SAF.

Data collection for pregnancy, pregnancy outcomes, including congenital malformations, spontaneous abortion, elective abortion, stillbirth, ectopic pregnancy, molar pregnancy, and other important health conditions in the offspring is a secondary endpoint of the PREMIERE registry with its dedicated questionnaire.

The number of subjects with pregnancy, treatment status at start of pregnancy, number of pregnancy and outcomes will be presented by treatment group together and split by female subjects and for male participant pregnancy of partner.

Treatment status at start of pregnancy will be summarized as follows:

- <= 6 months after end of treatment: defined as start of pregnancy <= last dose + 183 days
- > 6 months after end of treatment: defined as start of pregnancy > last dose + 183 days

For start of pregnancy, the first date of the last menstrual period will be used. If this date is missing or partial, the estimated delivery date will be considered (minus 280 days for duration of pregnancy). If that estimated delivery date is also missing, the date of baby birth and gestational age at birth will be considered.

Descriptive statistics will be presented for the time (in days) from last dose to start of pregnancy for subjects who started pregnancy <= 6 months after end of treatment.

Mode of delivery, major delivery complication (y, n), infant child status (alive, deceased) and birth defects (y, n) will be presented.

A listing of AE related to pregnancy and a listing of pregnancy details will be presented.

All datasets with event collection of pregnancy, dedicated CRF pages or AE reporting or any other datasets will be considered as source of information. When information is taken from AE panels, all PTs from MedDRA SMQ (SMQ 20000185) labelled "SMQ 20000185 Pregnancy and neonatal topics" are identified (see Appendix 18.1). The obtained list is reviewed, and a decision is made for which events qualify as Pregnancies. These classifications are documented with reasons in Appendix 18.2 and read into the programs for calculations.

Note: the final list of AEs related to pregnancy may be revised after database lock. Any changes from the list above will be described in the CSR.

#### 15.3 Adverse Events

Reporting will be done for SAF.

Adverse events are events that are reported with a start date on or after the end of clinical trial + 1 day [Registry Day 1].

AEs collected in PREMIERE either from AEs CRF Pages (AE dataset) or New Diagnoses CRF Pages (CE dataset) will be included.

Seriousness is not collected for events in the New Diagnoses CRF Pages. Seriousness will not be imputed and therefore these diagnoses will not be included in serious or non-serious AE tables.

#### 15.3.1 All Adverse Events

All adverse events will be summarized following statistics described in section 15.1.1.

## Clinical trial.gov and EudraCT -requirements

In addition, a summary table will be provided for non-serious adverse events by SOC and PT per treatment group excluding SAEs applying

• frequency threshold of 5% based on crude incidence in either group

#### 15.3.2 Serious Adverse Events

Serious adverse events will be presented following statistics described in section 15.1.1

#### Clinical trial.gov and EudraCT -requirements

In addition, a summary table will be provided for serious adverse events by SOC and PT per treatment group.

## 15.4 Deaths, Other Serious Adverse Events, and Other Significant Adverse Events

#### **15.4.1 Deaths**

Adverse events leading to death will be presented following statistics described in section 15.1.1.

## 15.5 Adverse Event of Special Interest

The term Adverse Events of Special Interest represents a broader than usual category of events for which specific attention will be paid during the review of the results.

The following statistics will be presented:

• Summary: Patient-year, number of unique event, number of subjects with at least one event, crude incidence and 95% CI per treatment group. All these statistics will be repeated for AE leading to death and serious AE.

In addition, summary table will be repeated by

- o CLARITY only
- CLARITY/CLARITY EXTENSION
- o ORACLE MS
- o ONWARD
- By PT: Number of patients with the AE and crude incidence (%) per treatment group and total will be presented.

#### 15.5.1 **AESI= Infections**

Reporting will be regrouped into the 7 following AESI categories.

• AESI = Infections and Infestations

AESI = Infections and infestations is defined by any event belonging to the MedDRA SOC = Infections and Infestations.

• AESI = Severe Infections

AESI = Severe Infections is a custom grouping defined by any serious or severe event belonging to the MedDRA SOC = Infections and Infestations.

#### **Data Handling**

Adverse events collected under the New Diagnosis pages (PREMIERE eCRF only) does not have characteristics for severity being collected. However, AEs collected under the category "Other **severe** infections" will be considered for the definition of the AESI = Severe Infections.

• AESI = Herpetic infections

AESI = Herpetic infections is a custom grouping defined by any events from MedDRA HLT = Herpes viral infections.

• AESI = Opportunistic infections

The medical concept "opportunistic infections (including tuberculosis and PML)" is a custom grouping based on medical assessment. It includes MedDRA Preferred Terms (PTs) associated to viral, protozoal and bacterial infections as well as PTs associated to fungal infections with the exclusion of mucocutaneous and cutaneous fungal infections. Infections as provided by the US Centers of Disease Control (1993 revision) and in the Guidelines for the Prevention and Treatment of Opportunistic Infections in HIV-Infected Adults and Adolescents, http://aidsinfo.nih.gov/guidelines are included. PTs pertaining to the HLT 'Herpes viral infections' are not included.

This definition will be shortened in the tables footnote to read:

AESI = Opportunistic Infections is based on respective lists available in the context of HIV infections. It includes MedDRA preferred terms (PTs) associated to viral, fungal, protozoal and bacterial infections. PTs pertaining to the HLT 'Herpes viral infections' are not included.

The MedDRA terms that will be selected are listed in Appendix 18.3.

• AESI = Herpes zoster infections

AESI = Herpes zoster infections is a custom grouping defined by PTs with the term 'herpes zoster'.

The PTs that will be selected are listed in Appendix 18.4.

AESI = PML

AESI = PML is a custom grouping defined by any events from MedDRA HLT = Polyomavirus infection.

AESI = Tuberculosis

AESI = Tuberculosis is a custom grouping defined by any events from MedDRA HLT = Tuberculous infections.

## **15.5.2 AESI = Malignancies**

The AESI Malignancies is a custom query using the following process:

All PTs from MedDRA SMQ (SMQ code 20000091) labelled "Malignant or unspecified tumours" are identified (see Appendix 18.5). For this SMQ, there are no broad terms available. The obtained list is reviewed, and an adjudicated decision is made with documented justifications which events qualify as malignancies. These classifications are documented with reasons in Appendix 18.6 and read into the programs for calculations.

# 15.6 Handling of Missing or Partial AE Dates (onset, resolution date)

Incomplete AE-related dates will be handled in a 'worst case' manner to ensure no under-estimation of the duration of adverse events:

Onset date of an AE

- If the onset date of an AE is missing completely, or missing partially, but the onset month and year (or the onset year) is equal to Registry Day 1, then the onset date will be replaced by the minimum of Registry Day 1 and AE resolution date. Therefore, the period used for defining TEAEs is not underestimated.
- In all other cases, the missing onset day or missing onset month will be replaced by 1/January, ensuring that no adverse event duration is under-estimated.

Stop date of an AE

- Incomplete stop dates will be replaced by the last day of the month (if day is missing), and December (if the month is missing), unless resulting in a date later than the date of subject's death. In the latter case, the date of death will be used to impute the incomplete stop date.
- In all other cases, (for example where the day and month are missing) the incomplete stop date will not be imputed.

## 15.7 Clinical Laboratory Evaluation

Please refer to section 15.1.4.

## 15.8 Vital Signs

Not Applicable.

## 15.9 Other Safety or Tolerability Evaluations

Not Applicable.

#### 16 **Analyses of Other Endpoints**

Not Applicable.

#### 17 References

- 1. Clinical Study Report. EMR700568-012 Prospective observational long-term safety REgistry of Multiple sclerosis patients who have participated in cladribine clinical studies (PREMIERE). Merck KGaA, Darmstadt, Germany and in USA: EMD Serono, Inc., Rockland MA, USA. May 2 2016
- 2. Clinical Study Report. EMR700568-012 Prospective observational long-term safety registry of Multiple Sclerosis patients who have participated in cladribine clinical trials (PREMIERE). Merck Serono SA – Geneva An affiliate of Merck KGaA, Darmstadt, Germany, 29 quai des Bergues, 1201 Geneva / Switzerland. February 5 2018
- Clopper, C.J., and Pearson, E.S. The Use of Confidence or Fiducial Limits Illustrated in 3. the Case of the Binomial", (1934), "Biometrika 26, 404–41
- Jiming Fang Institute for Clinical Evaluative Sciences, Canada, 2011, Using SAS® 4. Procedures FREQ, GENMOD, LOGISTIC, and PHREG to Estimate Adjusted Relative Risks – A Case Study, Statistics and Data analysis, SAS Global Forum 2011.
- 5. Agresti, A., and Coull, B. (1998). Approximate is better than 'exact' for interval estimation of binomial proportions. The American Statistician, 52, 119-126.
- 6. Miettinen O, Nurminen M. Comparative analysis of two rates. Statistics in Medicine 1985; 4:213 -226
- 7. Common Terminology Criteria for Adverse Events v3.0 (CTCAE), Published August 9, 2006,

(https://ctep.cancer.gov/protocoldevelopment/electronic applications/docs/ctcaev3.pdf

## 18 Appendices

## 18.1 Pregnancy and neonatal topics (SMQ 20000185)


| Biotinidase deficiency 10071434 PT | |
|-----------------------------------------------------------------|---|
| Birth mark 10004950 PT | • |
| Birt-Hogg-Dube syndrome 10067736 PT | • |
| Bladder agenesis 10056655 PT | |
| Blau syndrome 10071755 PT | |
| Blepharophimosis congenital 10049241 PT | |
| Blindness congenital 10005176 PT | |
| Bloch-Sulzberger syndrome 10077624 PT | |
| Blood incompatibility haemolytic anaemia of newborn 10056369 PT | |
| Bloom syndrome 10073032 PT | |
| Brachycephaly 10053682 PT | |
| Brachydactyly 10072883 PT | |
| Brain malformation 10048409 PT | |
| Branchial cleft sinus 10006162 PT | |
| Branchial cyst 10006164 PT | |
| Branchiogenic syndrome 10058169 PT | |
| Branchio-oto-renal syndrome 10071135 PT | |
| Breast malformation 10006271 PT | |
| Bronchogenic cyst 10064585 PT | |
| Bruton's agammaglobulinaemia 10060360 PT | |
| Bulbospinal muscular atrophy congenital 10068597 PT | |
| Buried penis syndrome 10067131 PT | |
| Camptodactyly congenital 10049028 PT | |
| Camptomelia 10078297 PT | |
| Canavan disease 10067608 PT | |
| Cancer gene carrier 10052648 PT | |
| CANDLE syndrome 10073960 PT | |
| Carbamoyl phosphate synthetase deficiency 10058297 PT | |
| Carbohydrate metabolism disorder 10061023 PT | |
| Carcinogenic effect in offspring 10007268 PT | • |
| Cardiac lymphangioma 10055010 PT | • |
| Cardiac malposition 10007585 PT | |
| Cardiac septal defect 10064021 PT | • |
| Carney complex 10076601 PT | |
| Carnitine palmitoyltransferase deficiency 10050215 PT | • |
| Carnitine-acylcarnitine translocase deficiency 10078729 PT | |
| Carpus curvus 10007700 PT | |
| Cartilage-hair hypoplasia 10069596 PT | • |
| Cataract congenital 10007747 PT | • |
| Caudal regression syndrome 10059387 PT | • |
| Central core disease 10057620 PT | • |
| Central nervous system dermoid tumour 10007942 PT | • |
| Cerebellar dysplasia 10072942 PT | |
| Cerebellar hypoplasia 10008033 PT | |
| Cerebral arteriovenous malformation haemorrhagic 10008086 PT | |


| Endocardial fibroelastosis 10014663 PT Enteric duplication 10076653 PT Entropion congenital 10014923 PT Epidermal naevus 10014985 PT Epidermal naevus syndrome 10077952 PT Epidermolysis 10053177 PT Epidermolysis bullosa 10014989 PT Epilepsy congenital 10015039 PT Epispadias 10015088 PT Erythroblastosis foetalis 10015088 PT Erythrokeratodermia variabilis 10015487 PT Essential fructosuria 10015487 PT Exomphalos 10015677 PT Exomphalos 10015677 PT External auditory canal atresia 10054875 PT External auditory canal atresia 10072727 PT Eye anterior chamber congenital anomaly 10072727 PT Eyelid ptosis congenital 10015996 PT Fabry's disease 10016016 PT Factiony's disease 10016 |
|---|
| Entropion congenital 10014923 PT Epidermal naevus 10014985 PT Epidermal naevus syndrome 10077952 PT Epidermolysis 10053177 PT Epidermolysis bullosa 10014989 PT Epilepsy congenital 10015039 PT Epispadias 10015088 PT Erythroblastosis foetalis 10015251 PT Erythrokeratodermia variabilis 10015487 PT Exsential fructosuria 10015487 PT Exomphalos 10015487 PT Exophthalmos congenital 10050696 PT External auditory canal atresia 10054875 PT External pelvis 10072727 PT Eyel anterior chamber congenital anomaly 10015096 PT Eyelid ptosis congenital 10015996 PT Faciority disease 10016015 PT Faciority disease 10016016 PT Facioscapulohumeral muscular dystrophy 10064087 PT Factor II deficiency |
| Epidermal naevus 10014985 PT Epidermal naevus syndrome 10077952 PT Epidermolysis 10053177 PT Epidermolysis bullosa 10014989 PT Epilepsy congenital 10015003 PT Epispadias 10015088 PT Erythroblastosis foetalis 10015081 PT Erythrokeratodermia variabilis 10049048 PT Essential fructosuria 10015487 PT Exomphalos 10015677 PT Exophthalmos congenital 1005696 PT External auditory canal atresia 10054875 PT Extrarenal pelvis 10072727 PT Eye anterior chamber congenital anomaly 10061051 PT Eyelid ptosis congenital 10015096 PT Fabry's disease 10016016 PT Facioral I deficiency 1006071 PT Factor I deficiency 10016076 PT Factor III deficiency 10016076 PT Factor V Leiden carrier 1004893 |
| Epidermal naevus syndrome 10077952 PT Epidermolysis 10053177 PT Epidermolysis bullosa 10014989 PT Epilepsy congenital 10015038 PT Epispadias 10015088 PT Erythrolastosis foetalis 10015251 PT Erythrokeratodermia variabilis 10049048 PT Essential fructosuria 10015487 PT Exomphalos 10015677 PT Exomphalos congenital 1005696 PT External auditory canal atresia 10054875 PT Extrarenal pelvis 10054875 PT Eye anterior chamber congenital anomaly 10061051 PT Eyelid ptosis congenital 10015096 PT Fabry's disease 10016016 PT Faciodigitogenital dysplasia 10067141 PT Factor I deficiency 10064087 PT Factor I deficiency 10016075 PT Factor III deficiency 10016076 PT Factor V Leiden carrier <td< td=""></td<> |
| Epidermolysis 10053177 PT Epidermolysis bullosa 10014989 PT Epilepsy congenital 10015039 PT Epispadias 10015088 PT Erythroblastosis foetalis 10015251 PT Erythrokeratodermia variabilis 10049048 PT Essential fructosuria 10015487 PT Exomphalos 10015677 PT Exophthalmos congenital 1005696 PT External auditory canal atresia 10054875 PT Extrarenal pelvis 10072277 PT Eyelid ptosis congenital 10061051 PT Eyelid ptosis congenital 10016075 PT Eyelid ptosis congenital 10016016 PT Faciorizagonilal dysplasia 10016016 PT Faciorizagonilal dysplasia 10067141 PT Factor I deficiency 10016075 PT Factor I deficiency 10016075 PT Factor II deficiency 10016075 PT Factor IV deficiency 1001607 |
| Epidermolysis bullosa 10014989 PT Epilepsy congenital 10015039 PT Epispadias 10015088 PT Erythroblastosis foetalis 10015251 PT Erythrokeratodermia variabilis 10049048 PT Essential fructosuria 10015487 PT Exomphalos 10015677 PT Exophthalmos congenital 10050696 PT External auditory canal atresia 10054875 PT Extrarenal pelvis 10072727 PT Eye anterior chamber congenital anomaly 10061051 PT Eyelid ptosis congenital 10015996 PT Epolity's disease 10016016 PT Faciodigitogenital dysplasia 1006016 PT Factor I deficiency 10016075 PT Factor I deficiency 10016075 PT Factor II mutation 100504087 PT Factor IX deficiency 10016077 PT Factor V Leiden carrier 10075652 PT Factor V Leiden mutation |
| Epilepsy congenital 10015039 PT Epispadias 10015088 PT Erythroblastosis foetalis 10015251 PT Erythrokeratodermia variabilis 10049048 PT Essential fructosuria 10015487 PT Exomphalos 10015677 PT Exophthalmos congenital 10050696 PT External auditory canal atresia 10054875 PT Extrarenal pelvis 10072727 PT Eye anterior chamber congenital anomaly 10061051 PT Eyelid ptosis congenital 10015996 PT Epolity's disease 10016016 PT Faciodigitogenital dysplasia 10016016 PT Factor I deficiency 10016075 PT Factor I deficiency 10016075 PT Factor III deficiency 10016076 PT Factor III deficiency 10052473 PT Factor V deficiency 10016077 PT Factor V Leiden carrier 10075652 PT Factor V Leiden mutation |
| Epispadias 10015088 PT Erythroblastosis foetalis 10015251 PT Erythrokeratodermia variabilis 10049048 PT Essential fructosuria 10015487 PT Exomphalos 10015677 PT Exophthalmos congenital 10050696 PT External auditory canal atresia 10054875 PT Extrarenal pelvis 10072727 PT Eye anterior chamber congenital anomaly 10061051 PT Eyelid ptosis congenital 10016096 PT Fabry's disease 10016016 PT Faciodigitogenital dysplasia 10061051 PT Facioscapulohumeral muscular dystrophy 10064087 PT Factor I deficiency 10016075 PT Factor III deficiency 10016076 PT Factor III deficiency 10052473 PT Factor V Leiden carrier 10052473 PT Factor V Leiden mutation 10058279 PT Factor V Leiden mutation 1005609 PT Fact |
| Erythroblastosis foetalis 10015251 PT Erythrokeratodermia variabilis 10049048 PT Essential fructosuria 10015487 PT Exomphalos 10015677 PT Exophthalmos congenital 10050696 PT External auditory canal atresia 10054875 PT Extrarenal pelvis 10072727 PT Eye anterior chamber congenital anomaly 10061051 PT Eyeli ptosis congenital 10016096 PT Fabry's disease 10016016 PT Faciodigitogenital dysplasia 10061014 PT Facioscapulohumeral muscular dystrophy 10064087 PT Factor I deficiency 10016075 PT Factor III deficiency 10016076 PT Factor III deficiency 10052473 PT Factor V deficiency 10016077 PT Factor V Leiden carrier 10075652 PT Factor V Leiden mutation 10058279 PT Factor V Leiden mutation 10016080 PT |
| Erythrokeratodermia variabilis 10049048 PT Essential fructosuria 10015487 PT Exomphalos 10015677 PT Exophthalmos congenital 10050696 PT External auditory canal atresia 10054875 PT Extrarenal pelvis 10072727 PT Eye anterior chamber congenital anomaly 10061051 PT Eyelid ptosis congenital 10015996 PT Fabry's disease 10016016 PT Faciodigitogenital dysplasia 10067141 PT Facioscapulohumeral muscular dystrophy 10064087 PT Factor I deficiency 10016075 PT Factor II deficiency 10016075 PT Factor III deficiency 10055003 PT Factor IX deficiency 10016077 PT Factor V deficiency 10048930 PT Factor V Leiden carrier 10075652 PT Factor V Leiden mutation 10058279 PT Factor VIII deficiency 10016080 PT Fa |
| Essential fructosuria 10015487 PT Exomphalos 10015677 PT Exophthalmos congenital 10050696 PT External auditory canal atresia 10054875 PT Extrarenal pelvis 10072727 PT Eye anterior chamber congenital anomaly 10061051 PT Eyelid ptosis congenital 10015996 PT Fabry's disease 10016016 PT Faciodigitogenital dysplasia 10067141 PT Facioscapulohumeral muscular dystrophy 10064087 PT Factor I deficiency 10016075 PT Factor III deficiency 10016076 PT Factor III mutation 10052473 PT Factor IX deficiency 10016077 PT Factor V deficiency 10048930 PT Factor V Leiden carrier 10075652 PT Factor V Leiden mutation 10058279 PT Factor VIII deficiency 10016080 PT Factor VIII deficiency 10016080 PT Factor VIII deficiency 10016080 PT Factor X deficienc |
| Exomphalos 10015677 PT Exophthalmos congenital 10050696 PT External auditory canal atresia 10054875 PT Extrarenal pelvis 10072727 PT Eye anterior chamber congenital anomaly 10061051 PT Eyelid ptosis congenital 10015996 PT Fabry's disease 10016016 PT Faciodigitogenital dysplasia 10067141 PT Facioscapulohumeral muscular dystrophy 10064087 PT Factor I deficiency 10016075 PT Factor II deficiency 10016076 PT Factor III deficiency 10052473 PT Factor IX deficiency 10016077 PT Factor V deficiency 10048930 PT Factor V Leiden carrier 10075652 PT Factor VII deficiency 10016079 PT Factor VIII deficiency 10016080 PT Factor VIII deficiency 10016080 PT Factor X deficiency 10016080 PT |
| Exophthalmos congenital 10050696 PT External auditory canal atresia 10054875 PT Extrarenal pelvis 10072727 PT Eye anterior chamber congenital anomaly 10061051 PT Eyelid ptosis congenital 10015996 PT Fabry's disease 10016016 PT Faciodigitogenital dysplasia 10067141 PT Facioscapulohumeral muscular dystrophy 10064087 PT Factor I deficiency 10016075 PT Factor II deficiency 10016076 PT Factor III deficiency 10052473 PT Factor IX deficiency 10016077 PT Factor V deficiency 10048930 PT Factor V Leiden carrier 10075652 PT Factor VI Leiden mutation 10058279 PT Factor VIII deficiency 10016080 PT Factor VIII deficiency 10016080 PT Factor VIII deficiency 10016080 PT Factor VIII deficiency 10016080 PT |
| External auditory canal atresia 10054875 PT Extrarenal pelvis 10072727 PT Eye anterior chamber congenital anomaly 10061051 PT Eyelid ptosis congenital 10015996 PT Fabry's disease 10016016 PT Faciodigitogenital dysplasia 10067141 PT Facioscapulohumeral muscular dystrophy 10064087 PT Factor I deficiency 10016075 PT Factor III deficiency 10016076 PT Factor III mutation 10052033 PT Factor III deficiency 10016077 PT Factor IX deficiency 10016077 PT Factor V deficiency 10048930 PT Factor V Leiden carrier 10075652 PT Factor V Leiden mutation 10058279 PT Factor VIII deficiency 10016079 PT Factor VIII deficiency 10016080 PT Factor X deficiency 10016080 PT |
| Extrarenal pelvis 10072727 PT Eye anterior chamber congenital anomaly 10061051 PT Eyelid ptosis congenital 10015996 PT Fabry's disease 10016016 PT Faciodigitogenital dysplasia 10067141 PT Facioscapulohumeral muscular dystrophy 10064087 PT Factor I deficiency 10016075 PT Factor III deficiency 10016076 PT Factor III deficiency 10052473 PT Factor III deficiency 10016077 PT Factor IX deficiency 10016077 PT Factor V deficiency 10075652 PT Factor V Leiden carrier 10075652 PT Factor V Leiden mutation 10058279 PT Factor VIII deficiency 10016079 PT Factor VIII deficiency 10016079 PT Factor VIII deficiency 10016079 PT Factor VIII deficiency 10016079 PT Factor VIII deficiency 10016080 PT Factor VIII deficiency 10016080 PT Factor VIII deficiency 10016080 PT Factor V III deficiency 10016080 PT |
| Eye anterior chamber congenital anomaly10061051PTEyelid ptosis congenital10015996PTFabry's disease10016016PTFaciodigitogenital dysplasia10067141PTFacioscapulohumeral muscular dystrophy10064087PTFactor I deficiency10016075PTFactor III mutation10065003PTFactor III deficiency10052473PTFactor IX deficiency10016077PTFactor V deficiency10048930PTFactor V Leiden carrier10075652PTFactor V Leiden mutation10058279PTFactor VIII deficiency10016079PTFactor VIII deficiency10016079PTFactor VIII deficiency10016080PTFactor X deficiency10016080PTFactor X deficiency10052474PT |
| Eyelid ptosis congenital 10015996 PT Fabry's disease 10016016 PT Faciodigitogenital dysplasia 10067141 PT Facioscapulohumeral muscular dystrophy 10064087 PT Factor I deficiency 10016075 PT Factor III deficiency 10016076 PT Factor III deficiency 1005203 PT Factor IX deficiency 10016077 PT Factor V deficiency 10048930 PT Factor V Leiden carrier 10075652 PT Factor V Leiden mutation 10058279 PT Factor VIII deficiency 10016079 PT Factor VIII deficiency 10016080 PT Factor X deficiency 10052474 PT |
| Fabry's disease 10016016 PT Faciodigitogenital dysplasia 10067141 PT Facioscapulohumeral muscular dystrophy 10064087 PT Factor I deficiency 10016075 PT Factor II deficiency 10016076 PT Factor III mutation 10065003 PT Factor III deficiency 10016077 PT Factor IX deficiency 10016077 PT Factor V deficiency 10048930 PT Factor V Leiden carrier 10075652 PT Factor V Leiden mutation 10058279 PT Factor VIII deficiency 10016079 PT Factor VIII deficiency 10016079 PT Factor VIII deficiency 10016080 PT Factor X deficiency 10052474 PT |
| Faciodigitogenital dysplasia Facioscapulohumeral muscular dystrophy Factor I deficiency Factor II deficiency Factor III mutation Factor III deficiency Factor III deficiency Factor IX deficiency Factor V deficiency Factor V Leiden carrier Factor V Leiden mutation Factor VIII deficiency Factor VIII deficiency Factor V Leiden factor V |
| Facioscapulohumeral muscular dystrophy Factor I deficiency Factor II deficiency Factor III deficiency Factor III mutation Factor III deficiency Factor IX deficiency Factor IX deficiency Factor V deficiency Factor V Leiden carrier Factor V Leiden mutation Factor VII deficiency Factor V Leiden factor V Leiden mutation Factor VIII deficiency Factor V Leiden factor V Leiden mutation Factor VIII deficiency Factor VIII deficiency Factor VIII deficiency Factor VIII deficiency Factor V Leiden factor V Leiden factor V Leiden mutation Factor VIII deficiency Factor V Leiden factor V Leiden fact |
| Factor I deficiency 10016075 PT Factor II deficiency 10016076 PT Factor III mutation 10065003 PT Factor III deficiency 10052473 PT Factor IX deficiency 10016077 PT Factor V deficiency 10048930 PT Factor V Leiden carrier 10075652 PT Factor V Leiden mutation 10058279 PT Factor VIII deficiency 10016079 PT Factor VIII deficiency 10016080 PT Factor X deficiency 10052474 PT |
| Factor II deficiency 10016076 PT Factor II mutation 10065003 PT Factor III deficiency 10052473 PT Factor IX deficiency 10016077 PT Factor V deficiency 10048930 PT Factor V Leiden carrier 10075652 PT Factor V Leiden mutation 10058279 PT Factor VIII deficiency 10016079 PT Factor VIII deficiency 10016080 PT Factor X deficiency 10052474 PT |
| Factor II mutation 10065003 PT Factor III deficiency 10052473 PT Factor IX deficiency 10016077 PT Factor V deficiency 10048930 PT Factor V Leiden carrier 10075652 PT Factor V Leiden mutation 10058279 PT Factor VIII deficiency 10016079 PT Factor VIII deficiency 10016080 PT Factor X deficiency 10052474 PT |
| Factor III deficiency 10052473 PT Factor IX deficiency 10016077 PT Factor V deficiency 10048930 PT Factor V Leiden carrier 10075652 PT Factor V Leiden mutation 10058279 PT Factor VII deficiency 10016079 PT Factor VIII deficiency 10016080 PT Factor X deficiency 10052474 PT |
| Factor IX deficiency 10016077 PT Factor V deficiency 10048930 PT Factor V Leiden carrier 10075652 PT Factor V Leiden mutation 10058279 PT Factor VII deficiency 10016079 PT Factor VIII deficiency 10016080 PT Factor X deficiency 10052474 PT |
| Factor V deficiency 10048930 PT Factor V Leiden carrier 10075652 PT Factor V Leiden mutation 10058279 PT Factor VII deficiency 10016079 PT Factor VIII deficiency 10016080 PT Factor X deficiency 10052474 PT |
| Factor V Leiden carrier Factor V Leiden mutation Factor VII deficiency Factor VIII deficiency Factor X deficiency Factor X deficiency 10075652 PT |
| Factor V Leiden mutation 10058279 PT Factor VII deficiency 10016079 PT Factor VIII deficiency 10016080 PT Factor X deficiency 10052474 PT |
| Factor VII deficiency 10016079 PT Factor VIII deficiency 10016080 PT Factor X deficiency 10052474 PT |
| Factor VIII deficiency 10016080 PT Factor X deficiency 10052474 PT |
| Factor X deficiency 10052474 PT |
| • |
| Factor XI deficiency 10016082 PT |
| Factor XII deficiency 10051806 PT |
| Factor XIII deficiency 10016083 PT |
| Fallot's pentalogy 10059205 PT |
| Fallot's tetralogy 10016193 PT |
| Fallot's trilogy 10064011 PT |
| Familial acromegaly 10080509 PT |
| Familial amyloidosis 10016202 PT |
| Familial amyotrophic lateral sclerosis 10077024 PT |
| Familial cold autoinflammatory syndrome 10064570 PT |
| Familial haemophagocytic lymphohistiocytosis 10070904 PT |
| Familial hemiplegic migraine 10067039 PT |
| Familial high density lipoprotein deficiency 10079119 PT |

| Familial hypertriglyceridaemia10059183PTFamilial hypocalciuric hypercalcaemia10068698PTFamilial infantile bilateral striatal necrosis10077450PTFamilial isolated hyperparathyroidism10080773PTFamilial mediterranean fever10016207PTFamilial medullary thyroid cancer10073153PTFamilial periodic paralysis10016208PTFamilial periodic paralysis10016209PTFamilial renal glycosuria10073689PTFamilial renal glycosuria10073689PTFamilial tremor10016212PTFamilial tremor10016212PTFatal familial insomnia10072077PTFatty acid oxidation disorder10077951PTFemoral anteversion10064516PTFemoral retroversion10064514PTFemur-fibula-ulna complex10068448PTFibrous dysplasia osificans progressiva10068448PTFibrous dysplasia of bone10016664PTFibrous dysplasia of jaw10070535PTFibula agenesis10054882PTFibula agenesis10054882PTFibula je-Harbor syndrome10079943PTFoetal alcohol syndrome10016845PTFoetal anticonvulsant syndrome10066485PT |
|---|
| Familial infantile bilateral striatal necrosis 10077450 PT Familial isolated hyperparathyroidism 10080773 PT Familial mediterranean fever 10016207 PT Familial medullary thyroid cancer 10073153 PT Familial periodic paralysis 10016208 PT Familial polycythaemia 10016209 PT Familial renal glycosuria 10073689 PT Familial tremor 10072229 PT Familial tremor 10016212 PT Fanconi syndrome 10016212 PT Fatal familial insomnia 10072077 PT Fatty acid oxidation disorder 10077951 PT Femoral anteversion 10064516 PT Femoral retroversion 10064516 PT Femur-fibula-ulna complex 10068448 PT Fibrous dysplasia ossificans progressiva 10068715 PT Fibrous dysplasia of bone 10016664 PT Fibula agenesis 10054882 PT Fibula agenesis 10016715 PT |
| Familial isolated hyperparathyroidism10080773PTFamilial mediterranean fever10016207PTFamilial medullary thyroid cancer10073153PTFamilial periodic paralysis10016208PTFamilial polycythaemia10016209PTFamilial renal glycosuria10073689PTFamilial scaphocephaly syndrome10072229PTFamilial tremor10016212PTFanconi syndrome10016212PTFatal familial insomnia10072077PTFatty acid oxidation disorder10077951PTFemoral anteversion10064516PTFemoral retroversion10064514PTFemur-fibula-ulna complex10068448PTFibrodysplasia ossificans progressiva10068715PTFibrous dysplasia of bone10016664PTFibrous dysplasia of jaw10070535PTFibula agenesis10054882PTFissure of tongue, congenital10016715PTFloating-Harbor syndrome10079943PTFoetal alcohol syndrome10016845PT |
| Familial mediterranean fever 10016207 PT Familial medullary thyroid cancer 10073153 PT Familial periodic paralysis 10016208 PT Familial polycythaemia 10016209 PT Familial renal glycosuria 10073689 PT Familial tremor 10072229 PT Familial tremor 10016212 PT Fanconi syndrome 10016212 PT Fatal familial insomnia 10072077 PT Fatty acid oxidation disorder 10077951 PT Femoral anteversion 10064516 PT Femoral retroversion 10064514 PT Femur-fibula-ulna complex 10068448 PT Fibrodysplasia ossificans progressiva 10068715 PT Fibrous dysplasia of bone 10016664 PT Fibrous dysplasia of jaw 10070535 PT Fibula agenesis 10054882 PT Fisure of tongue, congenital 10016715 PT Floating-Harbor syndrome 10079943 PT |
| Familial medullary thyroid cancer10073153PTFamilial periodic paralysis10016208PTFamilial polycythaemia10016209PTFamilial renal glycosuria10073689PTFamilial scaphocephaly syndrome10072229PTFamilial tremor10016212PTFanconi syndrome10016219PTFatal familial insomnia10072077PTFatty acid oxidation disorder10077951PTFemoral anteversion10064516PTFemoral retroversion10064514PTFemur-fibula-ulna complex10068448PTFibrodysplasia ossificans progressiva10068448PTFibrous dysplasia of bone10016664PTFibrous dysplasia of jaw10070535PTFibula agenesis10054882PTFissure of tongue, congenital10016715PTFloating-Harbor syndrome10079943PTFoetal alcohol syndrome10076845PT |
| Familial periodic paralysis10016208PTFamilial polycythaemia10016209PTFamilial renal glycosuria10073689PTFamilial scaphocephaly syndrome10072229PTFamilial tremor10016212PTFanconi syndrome10016219PTFatal familial insomnia10072077PTFatty acid oxidation disorder10077951PTFemoral anteversion10064516PTFemoral retroversion10064514PTFemur-fibula-ulna complex10068448PTFibrodysplasia ossificans progressiva10016664PTFibrous dysplasia of bone10016664PTFibrous dysplasia of jaw10070535PTFibula agenesis10054882PTFissure of tongue, congenital10016715PTFloating-Harbor syndrome10079943PTFoetal alcohol syndrome10016845PT |
| Familial polycythaemia10016209PTFamilial renal glycosuria10073689PTFamilial scaphocephaly syndrome10072229PTFamilial tremor10016212PTFanconi syndrome10016219PTFatal familial insomnia10072077PTFatty acid oxidation disorder10077951PTFemoral anteversion10064516PTFemoral retroversion10064514PTFemur-fibula-ulna complex10068448PTFibrodysplasia ossificans progressiva10068715PTFibrous dysplasia of bone10016664PTFibrous dysplasia of jaw10070535PTFibula agenesis10054882PTFissure of tongue, congenital10016715PTFloating-Harbor syndrome10079943PTFoetal alcohol syndrome10016845PT |
| Familial renal glycosuria10073689PTFamilial scaphocephaly syndrome10072229PTFamilial tremor10016212PTFanconi syndrome10016219PTFatal familial insomnia10072077PTFatty acid oxidation disorder10077951PTFemoral anteversion10064516PTFemoral retroversion10064514PTFemur-fibula-ulna complex10068448PTFibrodysplasia ossificans progressiva10068715PTFibrous dysplasia of bone10016664PTFibrous dysplasia of jaw10070535PTFibula agenesis10054882PTFissure of tongue, congenital10016715PTFloating-Harbor syndrome10079943PTFoetal alcohol syndrome10016845PT |
| Familial scaphocephaly syndrome Familial tremor Familial tremor Fanconi syndrome 10016212 FT Fanconi syndrome 10016219 FT Fatal familial insomnia 10072077 FT Fatty acid oxidation disorder 10077951 FT Femoral anteversion 10064516 FT Femoral retroversion 10064514 FT Femur-fibula-ulna complex 10068448 FT Fibrodysplasia ossificans progressiva 10068715 FT Fibrous dysplasia of bone 10016664 FT Fibrous dysplasia of jaw 10070535 FT Fibula agenesis 10054882 FT Fissure of tongue, congenital Floating-Harbor syndrome 10079943 FT Foetal alcohol syndrome |
| Familial tremor10016212PTFanconi syndrome10016219PTFatal familial insomnia10072077PTFatty acid oxidation disorder10077951PTFemoral anteversion10064516PTFemoral retroversion10064514PTFemur-fibula-ulna complex10068448PTFibrodysplasia ossificans progressiva10068715PTFibrous dysplasia of bone10016664PTFibrous dysplasia of jaw10070535PTFibula agenesis10054882PTFissure of tongue, congenital10016715PTFloating-Harbor syndrome10079943PTFoetal alcohol syndrome10016845PT |
| Fanconi syndrome10016219PTFatal familial insomnia10072077PTFatty acid oxidation disorder10077951PTFemoral anteversion10064516PTFemoral retroversion10064514PTFemur-fibula-ulna complex10068448PTFibrodysplasia ossificans progressiva10068715PTFibrous dysplasia of bone10016664PTFibrous dysplasia of jaw10070535PTFibula agenesis10054882PTFissure of tongue, congenital10016715PTFloating-Harbor syndrome10079943PTFoetal alcohol syndrome10016845PT |
| Fatal familial insomnia 10072077 PT Fatty acid oxidation disorder 10077951 PT Femoral anteversion 10064516 PT Femoral retroversion 10064514 PT Femur-fibula-ulna complex 10068448 PT Fibrodysplasia ossificans progressiva 10068715 PT Fibrous dysplasia of bone 10016664 PT Fibrous dysplasia of jaw 10070535 PT Fibula agenesis 10054882 PT Fissure of tongue, congenital 10016715 PT Floating-Harbor syndrome 10079943 PT Foetal alcohol syndrome 10016845 PT |
| Fatty acid oxidation disorder Femoral anteversion Femoral retroversion Femur-fibula-ulna complex Fibrodysplasia ossificans progressiva Fibrous dysplasia of bone Fibrous dysplasia of jaw Fibrous dy |
| Femoral anteversion10064516PTFemoral retroversion10064514PTFemur-fibula-ulna complex10068448PTFibrodysplasia ossificans progressiva10068715PTFibrous dysplasia of bone10016664PTFibrous dysplasia of jaw10070535PTFibula agenesis10054882PTFissure of tongue, congenital10016715PTFloating-Harbor syndrome10079943PTFoetal alcohol syndrome10016845PT |
| Femoral retroversion 10064514 PT Femur-fibula-ulna complex 10068448 PT Fibrodysplasia ossificans progressiva 10068715 PT Fibrous dysplasia of bone 10016664 PT Fibrous dysplasia of jaw 10070535 PT Fibula agenesis 10054882 PT Fissure of tongue, congenital 10016715 PT Floating-Harbor syndrome 10079943 PT Foetal alcohol syndrome 10016845 PT |
| Femur-fibula-ulna complex10068448PTFibrodysplasia ossificans progressiva10068715PTFibrous dysplasia of bone10016664PTFibrous dysplasia of jaw10070535PTFibula agenesis10054882PTFissure of tongue, congenital10016715PTFloating-Harbor syndrome10079943PTFoetal alcohol syndrome10016845PT |
| Fibrodysplasia ossificans progressiva 10068715 PT Fibrous dysplasia of bone 10016664 PT Fibrous dysplasia of jaw 10070535 PT Fibula agenesis 10054882 PT Fissure of tongue, congenital 10016715 PT Floating-Harbor syndrome 10079943 PT Foetal alcohol syndrome 10016845 PT |
| Fibrous dysplasia of bone 10016664 PT Fibrous dysplasia of jaw 10070535 PT Fibula agenesis 10054882 PT Fissure of tongue, congenital 10016715 PT Floating-Harbor syndrome 10079943 PT Foetal alcohol syndrome 10016845 PT |
| Fibrous dysplasia of jaw 10070535 PT Fibula agenesis 10054882 PT Fissure of tongue, congenital 10016715 PT Floating-Harbor syndrome 10079943 PT Foetal alcohol syndrome 10016845 PT |
| Fibula agenesis 10054882 PT Fissure of tongue, congenital 10016715 PT Floating-Harbor syndrome 10079943 PT Foetal alcohol syndrome 10016845 PT |
| Fissure of tongue, congenital 10016715 PT Floating-Harbor syndrome 10079943 PT Foetal alcohol syndrome 10016845 PT |
| Floating-Harbor syndrome 10079943 PT Foetal alcohol syndrome 10016845 PT |
| Foetal alcohol syndrome 10016845 PT |
| · |
| Foetal anticonvulsant syndrome 10066485 PT |
| Foetal chromosome abnormality 10064041 PT |
| Foetal cystic hygroma 10052011 PT |
| Foetal malformation 10060919 PT |
| Foetal megacystis 10073660 PT |
| Foetal methotrexate syndrome 10071183 PT |
| Foetal retinoid syndrome 10073720 PT |
| Foetal warfarin syndrome 10051445 PT |
| Foramen magnum stenosis 10064157 PT |
| Fragile X carrier 10052657 PT |
| Fragile X syndrome 10017324 PT |
| Fraser syndrome 10080219 PT |
| Frasier syndrome 10080313 PT |
| Freeman-Sheldon syndrome 10073655 PT |
| Frenulum breve 10072007 PT |
| Friedreich's ataxia 10017374 PT |
| Fryns syndrome 10075223 PT |
| Galactosaemia 10017604 PT |
| Gallbladder agenesis 10079018 PT |
| Gallbladder anomaly congenital 10061163 PT |
| Gastrointestinal arteriovenous malformation 10017932 PT |


| Retinal anomaly congenital 10038821 PT Retinal arteriovenous malformation 10038824 PT Retinal coloboma 10052643 PT Retinitis pigmentosa 10038914 PT Retinopathy congenital 10050706 PT Retinoschisis congenital 10038938 PT Rett syndrome 10077709 PT Rhesus haemolytic disease of newborn 10039037 PT Rib hypoplasia 10048893 PT Rib synostosis 10076624 PT Right aortic arch 10067407 PT Right ventricle outflow tract obstruction 10064195 PT Right ventricular false tendon 10080132 PT Right-to-left cardiac shunt 10076605 PT Riley-Day syndrome 10039179 PT Rippling muscle disease 10069417 PT Rotor's syndrome 10039234 PT Rubinstein-Taybi syndrome 10039281 PT Sacral hypoplasia 10064932 PT |
|---|
| Retinal coloboma 10052643 PT Retinitis pigmentosa 10038914 PT Retinopathy congenital 10050706 PT Retinoschisis congenital 10038938 PT Rett syndrome 10077709 PT Rhesus haemolytic disease of newborn 10039037 PT Rib hypoplasia 10048893 PT Rib synostosis 10076624 PT Right aortic arch 10067407 PT Right ventricle outflow tract obstruction 10064195 PT Right ventricular false tendon 10080132 PT Right-to-left cardiac shunt 10076605 PT Riley-Day syndrome 10039179 PT Rippling muscle disease 10069417 PT Rotor's syndrome 10039234 PT Rubinstein-Taybi syndrome 10039281 PT Sacral hypoplasia 10056659 PT |
| Retinitis pigmentosa10038914PTRetinopathy congenital10050706PTRetinoschisis congenital10038938PTRett syndrome10077709PTRhesus haemolytic disease of newborn10039037PTRib hypoplasia10048893PTRib synostosis10076624PTRight aortic arch10067407PTRight ventricle outflow tract obstruction10064195PTRight ventricular false tendon10080132PTRight-to-left cardiac shunt10076605PTRiley-Day syndrome10039179PTRippling muscle disease10069417PTRotor's syndrome10039234PTRubinstein-Taybi syndrome10039281PTSacral hypoplasia10056659PT |
| Retinopathy congenital10050706PTRetinoschisis congenital10038938PTRett syndrome10077709PTRhesus haemolytic disease of newborn10039037PTRib hypoplasia10048893PTRib synostosis10076624PTRight aortic arch10067407PTRight ventricle outflow tract obstruction10064195PTRight ventricular false tendon10080132PTRight-to-left cardiac shunt10076605PTRiley-Day syndrome10039179PTRippling muscle disease10069417PTRotor's syndrome10039234PTRubinstein-Taybi syndrome10039281PTSacral hypoplasia10056659PT |
| Retinoschisis congenital Rett syndrome 10038938 PT Rett syndrome 10077709 PT Rhesus haemolytic disease of newborn Rib hypoplasia 10048893 PT Rib synostosis 10076624 PT Right aortic arch 10067407 PT Right ventricle outflow tract obstruction 10064195 PT Right ventricular false tendon 10080132 PT Right-to-left cardiac shunt 10076605 PT Riley-Day syndrome 10039179 PT Rippling muscle disease 10069417 PT Rotor's syndrome 10039234 PT Rubinstein-Taybi syndrome 10039281 PT Sacral hypoplasia |
| Rett syndrome 10077709 PT Rhesus haemolytic disease of newborn 10039037 PT Rib hypoplasia 10048893 PT Rib synostosis 10076624 PT Right aortic arch 10067407 PT Right ventricle outflow tract obstruction 10064195 PT Right ventricular false tendon 10080132 PT Right-to-left cardiac shunt 10076605 PT Riley-Day syndrome 10039179 PT Rippling muscle disease 10069417 PT Rotor's syndrome 10039234 PT Rubinstein-Taybi syndrome 10039281 PT Sacral hypoplasia 10056659 PT |
| Rhesus haemolytic disease of newborn10039037PTRib hypoplasia10048893PTRib synostosis10076624PTRight aortic arch10067407PTRight ventricle outflow tract obstruction10064195PTRight ventricular false tendon10080132PTRight-to-left cardiac shunt10076605PTRiley-Day syndrome10039179PTRippling muscle disease10069417PTRotor's syndrome10039234PTRubinstein-Taybi syndrome10039281PTSacral hypoplasia10056659PT |
| Rib hypoplasia 10048893 PT Rib synostosis 10076624 PT Right aortic arch 10067407 PT Right ventricle outflow tract obstruction 10064195 PT Right ventricular false tendon 10080132 PT Right-to-left cardiac shunt 10076605 PT Riley-Day syndrome 10039179 PT Rippling muscle disease 10069417 PT Rotor's syndrome 10039234 PT Rubinstein-Taybi syndrome 10039281 PT Sacral hypoplasia 10056659 PT |
| Rib synostosis 10076624 PT Right aortic arch 10067407 PT Right ventricle outflow tract obstruction 10064195 PT Right ventricular false tendon 10080132 PT Right-to-left cardiac shunt 10076605 PT Riley-Day syndrome 10039179 PT Rippling muscle disease 10069417 PT Rotor's syndrome 10039234 PT Rubinstein-Taybi syndrome 10039281 PT Sacral hypoplasia 10056659 PT |
| Right aortic arch10067407PTRight ventricle outflow tract obstruction10064195PTRight ventricular false tendon10080132PTRight-to-left cardiac shunt10076605PTRiley-Day syndrome10039179PTRippling muscle disease10069417PTRotor's syndrome10039234PTRubinstein-Taybi syndrome10039281PTSacral hypoplasia10056659PT |
| Right ventricle outflow tract obstruction Right ventricular false tendon Right-to-left cardiac shunt Riley-Day syndrome Rippling muscle disease Rotor's syndrome Rubinstein-Taybi syndrome Sacral hypoplasia 10064195 PT 10080132 PT 10076605 PT 10039179 PT 10039234 PT 10039281 PT 10056659 PT |
| Right ventricular false tendon10080132PTRight-to-left cardiac shunt10076605PTRiley-Day syndrome10039179PTRippling muscle disease10069417PTRotor's syndrome10039234PTRubinstein-Taybi syndrome10039281PTSacral hypoplasia10056659PT |
| Right-to-left cardiac shunt 10076605 PT Riley-Day syndrome 10039179 PT Rippling muscle disease 10069417 PT Rotor's syndrome 10039234 PT Rubinstein-Taybi syndrome 10039281 PT Sacral hypoplasia 10056659 PT |
| Riley-Day syndrome 10039179 PT Rippling muscle disease 10069417 PT Rotor's syndrome 10039234 PT Rubinstein-Taybi syndrome 10039281 PT Sacral hypoplasia 10056659 PT |
| Rippling muscle disease 10069417 PT Rotor's syndrome 10039234 PT Rubinstein-Taybi syndrome 10039281 PT Sacral hypoplasia 10056659 PT |
| Rotor's syndrome10039234PTRubinstein-Taybi syndrome10039281PTSacral hypoplasia10056659PT |
| Rubinstein-Taybi syndrome 10039281 PT Sacral hypoplasia 10056659 PT |
| Sacral hypoplasia 10056659 PT |
| Sacralisation 10064932 PT |
| Sarcosinaemia 10059299 PT |
| Scaphocephaly 10049426 PT |
| Schimke immunoosseous dysplasia 10048699 PT |
| Schinzel-Giedion syndrome 10063540 PT |
| Schizencephaly 10073487 PT |
| Scimitar syndrome 10051951 PT |
| Sclerotylosis 10070504 PT |
| Sebaceous naevus 10039785 PT |
| Sensory neuropathy hereditary 10040037 PT |
| Septate hymen 10068484 PT |
| Septo-optic dysplasia 10067159 PT |
| Septum pellucidum agenesis 10062267 PT |
| Sertoli-cell-only syndrome 10066833 PT |
| Severe myoclonic epilepsy of infancy 10073677 PT |
| Sex chromosome abnormality 10061513 PT |
| Shawl scrotum 10080319 PT |
| Shone complex 10066802 PT |
| Short-chain acyl-coenzyme A dehydrogenase deficiency 10072655 PT |
| Shwachman-Diamond syndrome 10067940 PT |
| Sickle cell anaemia 10040641 PT |
| Sickle cell disease 10040644 PT |
| Sickle cell trait 10040650 PT |
| Silver-Russell syndrome 10062282 PT |
| Single umbilical artery 10049807 PT |
| Sirenomelia 10072457 PT |


| Oligohydramnios 10030289 PT Omphalorrhexis 10064270 PT Paternal exposure before pregnancy 10080093 PT Paternal exposure during pregnancy 10080092 PT Paternal exposure timing unspecified 10080092 PT Pelvic haematoma obstetric 10034248 PT Perineal repair breakdown 10034528 PT Peripartum cardiomyopathy 10049430 PT Peripartum haemorrhage 10072693 PT Placenta accreta 10062936 PT Placenta praevia 10035119 PT Placental praevia haemorrhage 10035119 PT Placental chorioangioma 10035112 PT Placental disorder 10035132 PT Placental disorder 10035132 PT Placental infarction 10068326 PT Placental insufficiency 10035138 PT Placental neoplasm 10064620 PT Placental polyp 10035142 PT Placental transfusi |
|---|
| Paternal exposure before pregnancy 10080093 PT Paternal exposure during pregnancy 10080091 PT Paternal exposure timing unspecified 10080092 PT Pelvic haematoma obstetric 10034248 PT Perineal repair breakdown 10034528 PT Peripartum cardiomyopathy 10049430 PT Peripartum haemorrhage 10072693 PT Placenta accreta 10062936 PT Placenta praevia 10035119 PT Placenta praevia haemorrhage 10035119 PT Placental praevia haemorrhage 10035121 PT Placental chorioangioma 10056718 PT Placental disorder 10035132 PT Placental dysplasia 1005471 PT Placental infarction 10068326 PT Placental infarction 10064620 PT Placental necrosis 10035138 PT Placental polyp 10035142 PT Placental polyp 10035142 PT Polymorp |
| Paternal exposure during pregnancy 10080091 PT Paternal exposure timing unspecified 10080092 PT Pelvic haematoma obstetric 10034248 PT Perineal repair breakdown 10034528 PT Peripartum cardiomyopathy 10049430 PT Peripartum haemorrhage 10072693 PT Placenta accreta 10062936 PT Placenta praevia 10035119 PT Placenta praevia haemorrhage 10035121 PT Placental chorioangioma 10056718 PT Placental disorder 10035132 PT Placental dysplasia 10054810 PT Placental hypertrophy 10068326 PT Placental infarction 1006420 PT Placental insufficiency 10035138 PT Placental necrosis 10035139 PT Placental neoplasm 10061349 PT Placental transfusion syndrome 10035142 PT Polymorphic eruption of pregnancy 10066100 PT |
| Paternal exposure timing unspecified 10080092 PT Pelvic haematoma obstetric 10034248 PT Perineal repair breakdown 10034528 PT Peripartum cardiomyopathy 10049430 PT Peripartum haemorrhage 10072693 PT Placenta accreta 10062936 PT Placenta praevia 10035119 PT Placenta praevia haemorrhage 10035121 PT Placental chorioangioma 10056718 PT Placental disorder 10035132 PT Placental disorder 10035132 PT Placental hypertrophy 10068326 PT Placental infarction 10068326 PT Placental necrosis 10035138 PT Placental necrosis 10035139 PT Placental neoplasm 10061349 PT Placental transfusion syndrome 10035142 PT Polyhydramnios 10035146 PT Polytpartum disorder 10066100 PT Postpartum haemorrhage |
| Pelvic haematoma obstetric 10034248 PT Perineal repair breakdown 10034528 PT Peripartum cardiomyopathy 10049430 PT Peripartum haemorrhage 10072693 PT Placenta accreta 10062936 PT Placenta praevia 10035119 PT Placenta praevia haemorrhage 10035121 PT Placental chorioangioma 10056718 PT Placental disorder 10035132 PT Placental disorder 10035132 PT Placental dysplasia 10054810 PT Placental hypertrophy 10068326 PT Placental infarction 10068326 PT Placental insufficiency 10035133 PT Placental necrosis 10035139 PT Placental neoplasm 10035139 PT Placental transfusion syndrome 10035142 PT Polyhydramnios 10036079 PT Polymorphic eruption of pregnancy 10066100 PT Postpartum haemorrhage |
| Perineal repair breakdown 10034528 PT Peripartum cardiomyopathy 10049430 PT Peripartum haemorrhage 10072693 PT Placenta accreta 10062936 PT Placenta praevia 10035119 PT Placenta praevia haemorrhage 10035121 PT Placental chorioangioma 10056718 PT Placental disorder 10035132 PT Placental dysplasia 10054810 PT Placental hypertrophy 10068326 PT Placental infarction 10064620 PT Placental infarction 10035138 PT Placental necrosis 10035139 PT Placental neoplasm 10035139 PT Placental polyp 10035146 PT Placental transfusion syndrome 10035146 PT Polyhydramnios 10036079 PT Polymorphic eruption of pregnancy 10066100 PT Postpartum haemorrhage 10036417 PT Postpartum hypopituitarism 10036419 PT Postpartum neurosis 10036419 PT Postpartum sepsis 10036422 PT |
| Peripartum cardiomyopathy 10049430 PT Peripartum haemorrhage 10072693 PT Placenta accreta 10062936 PT Placenta praevia 10035119 PT Placenta praevia haemorrhage 10035121 PT Placental chorioangioma 10056718 PT Placental disorder 10035132 PT Placental dysplasia 10054810 PT Placental hypertrophy 10068326 PT Placental infarction 10068326 PT Placental insufficiency 10035138 PT Placental necrosis 10035139 PT Placental neoplasm 10035139 PT Placental polyp 10035142 PT Placental transfusion syndrome 10035142 PT Polymorphic eruption of pregnancy 10036079 PT Postpartum haemorrhage 1006100 PT Postpartum hypopituitarism 10036417 PT Postpartum neurosis 10036419 PT Postpartum sepsis 10036422 PT |
| Peripartum haemorrhage 10072693 PT Placenta accreta 10062936 PT Placenta praevia 10035119 PT Placenta praevia haemorrhage 10035121 PT Placental chorioangioma 10056718 PT Placental disorder 10035132 PT Placental dysplasia 10054810 PT Placental hypertrophy 10068326 PT Placental infarction 10064620 PT Placental insufficiency 10035138 PT Placental necrosis 10035139 PT Placental neoplasm 10035139 PT Placental polyp 10035142 PT Placental transfusion syndrome 10035142 PT Polymorphic eruption of pregnancy 10036079 PT Postpartum disorder 1006100 PT Postpartum haemorrhage 10036417 PT Postpartum hypopituitarism 10036419 PT Postpartum neurosis 10036419 PT Postpartum sepsis 100364 |
| Placenta accreta 10062936 PT Placenta praevia 10035119 PT Placenta praevia haemorrhage 10035121 PT Placental chorioangioma 10056718 PT Placental disorder 10035132 PT Placental dysplasia 10054810 PT Placental hypertrophy 10068326 PT Placental infarction 10068326 PT Placental insufficiency 10035138 PT Placental necrosis 10035139 PT Placental neoplasm 10035139 PT Placental polyp 10035142 PT Placental transfusion syndrome 10035142 PT Polyhydramnios 10036079 PT Polymorphic eruption of pregnancy 1006100 PT Postpartum disorder 10061469 PT Postpartum hypopituitarism 10036417 PT Postpartum neurosis 10036419 PT Postpartum neurosis 10036419 PT Postpartum sepsis 10036422 |
| Placenta praevia 10035119 PT Placenta praevia haemorrhage 10035121 PT Placental chorioangioma 10056718 PT Placental disorder 10035132 PT Placental dysplasia 10054810 PT Placental hypertrophy 10068326 PT Placental infarction 10068326 PT Placental insufficiency 10035138 PT Placental necrosis 10035139 PT Placental neoplasm 10035139 PT Placental polyp 10035142 PT Placental transfusion syndrome 10035146 PT Polyhydramnios 10036079 PT Polymorphic eruption of pregnancy 1006100 PT Postpartum disorder 10061469 PT Postpartum hypopituitarism 10036417 PT Postpartum neurosis 10036419 PT Postpartum sepsis 10036422 PT |
| Placenta praevia haemorrhage Placental chorioangioma 10056718 PT Placental disorder 10035132 PT Placental dysplasia Placental hypertrophy 10068326 PT Placental infarction 10064620 PT Placental insufficiency 10035138 PT Placental necrosis 10035139 PT Placental neoplasm Placental neoplasm 10061349 PT Placental transfusion syndrome 10035142 PT Placental transfusion syndrome 10035146 PT Polyhydramnios 10036079 PT Postpartum disorder Postpartum haemorrhage 10036417 PT Postpartum hypopituitarism 10036419 PT Postpartum neurosis 10036419 PT Postpartum sepsis |
| Placental chorioangioma Placental disorder Placental disorder Placental dysplasia Placental hypertrophy Placental infarction Placental insufficiency Placental insufficiency Placental necrosis PT Placental neoplasm Placental neoplasm Placental polyp Placental transfusion syndrome Placental transfusion of pregnancy Polyhydramnios PT Postpartum disorder Postpartum hypopituitarism Postpartum neurosis PT Postpartum neurosis PT Postpartum sepsis PT Postpartum sepsis |
| Placental disorder10035132PTPlacental dysplasia10054810PTPlacental hypertrophy10068326PTPlacental infarction10064620PTPlacental insufficiency10035138PTPlacental necrosis10035139PTPlacental neoplasm10061349PTPlacental polyp10035142PTPlacental transfusion syndrome10035146PTPolyhydramnios10036079PTPolymorphic eruption of pregnancy10066100PTPostpartum disorder10036417PTPostpartum haemorrhage10036417PTPostpartum hypopituitarism10036419PTPostpartum neurosis10036419PTPostpartum sepsis10036422PT |
| Placental dysplasia10054810PTPlacental hypertrophy10068326PTPlacental infarction10064620PTPlacental insufficiency10035138PTPlacental necrosis10035139PTPlacental neoplasm10061349PTPlacental polyp10035142PTPlacental transfusion syndrome10035146PTPolyhydramnios10036079PTPolymorphic eruption of pregnancy10066100PTPostpartum disorder10061469PTPostpartum haemorrhage10036417PTPostpartum hypopituitarism10036297PTPostpartum neurosis10036419PTPostpartum sepsis10036422PT |
| Placental hypertrophy10068326PTPlacental infarction10064620PTPlacental insufficiency10035138PTPlacental necrosis10035139PTPlacental neoplasm10061349PTPlacental polyp10035142PTPlacental transfusion syndrome10035146PTPolyhydramnios10036079PTPolymorphic eruption of pregnancy10066100PTPostpartum disorder10061469PTPostpartum haemorrhage10036417PTPostpartum hypopituitarism10036297PTPostpartum neurosis10036419PTPostpartum sepsis10036422PT |
| Placental infarction10064620PTPlacental insufficiency10035138PTPlacental necrosis10035139PTPlacental neoplasm10061349PTPlacental polyp10035142PTPlacental transfusion syndrome10035146PTPolyhydramnios10036079PTPolymorphic eruption of pregnancy10066100PTPostpartum disorder10036419PTPostpartum haemorrhage10036417PTPostpartum hypopituitarism10036419PTPostpartum sepsis10036422PT |
| Placental insufficiency10035138PTPlacental necrosis10035139PTPlacental neoplasm10061349PTPlacental polyp10035142PTPlacental transfusion syndrome10035146PTPolyhydramnios10036079PTPolymorphic eruption of pregnancy10066100PTPostpartum disorder10061469PTPostpartum haemorrhage10036417PTPostpartum hypopituitarism10036297PTPostpartum neurosis10036419PTPostpartum sepsis10036422PT |
| Placental necrosis 10035139 PT Placental neoplasm 10061349 PT Placental polyp 10035142 PT Placental transfusion syndrome 10035146 PT Polyhydramnios 10036079 PT Polymorphic eruption of pregnancy 10066100 PT Postpartum disorder 10061469 PT Postpartum haemorrhage 10036417 PT Postpartum hypopituitarism 10036297 PT Postpartum neurosis 10036419 PT Postpartum sepsis 10036422 PT |
| Placental neoplasm Placental polyp Placental transfusion syndrome Polyhydramnios Polymorphic eruption of pregnancy Postpartum disorder Postpartum haemorrhage Postpartum hypopituitarism Postpartum neurosis Postpartum sepsis |
| Placental polyp10035142PTPlacental transfusion syndrome10035146PTPolyhydramnios10036079PTPolymorphic eruption of pregnancy10066100PTPostpartum disorder10061469PTPostpartum haemorrhage10036417PTPostpartum hypopituitarism10036297PTPostpartum neurosis10036419PTPostpartum sepsis10036422PT |
| Placental transfusion syndrome10035146PTPolyhydramnios10036079PTPolymorphic eruption of pregnancy10066100PTPostpartum disorder10061469PTPostpartum haemorrhage10036417PTPostpartum hypopituitarism10036297PTPostpartum neurosis10036419PTPostpartum sepsis10036422PT |
| Polyhydramnios10036079PTPolymorphic eruption of pregnancy10066100PTPostpartum disorder10061469PTPostpartum haemorrhage10036417PTPostpartum hypopituitarism10036297PTPostpartum neurosis10036419PTPostpartum sepsis10036422PT |
| Polymorphic eruption of pregnancy10066100PTPostpartum disorder10061469PTPostpartum haemorrhage10036417PTPostpartum hypopituitarism10036297PTPostpartum neurosis10036419PTPostpartum sepsis10036422PT |
| Postpartum disorder10061469PTPostpartum haemorrhage10036417PTPostpartum hypopituitarism10036297PTPostpartum neurosis10036419PTPostpartum sepsis10036422PT |
| Postpartum haemorrhage10036417PTPostpartum hypopituitarism10036297PTPostpartum neurosis10036419PTPostpartum sepsis10036422PT |
| Postpartum hypopituitarism10036297PTPostpartum neurosis10036419PTPostpartum sepsis10036422PT |
| Postpartum neurosis10036419PTPostpartum sepsis10036422PT |
| Postpartum sepsis 10036422 PT |
| and the second s |
| Postpartum stress disorder 10056394 PT |
| Postpartum thrombosis 10077022 PT |
| Postpartum uterine subinvolution 10036423 PT |
| Postpartum venous thrombosis 10036300 PT |
| Precipitate labour 10036519 PT |
| Pre-eclampsia 10036485 PT |
| Pregnancy in habitual aborter 10036562 PT |
| Pregnancy of unknown location 10072811 PT |
| Pregnancy with advanced maternal age 10036582 PT |
| Pregnancy with young maternal age 10069615 PT |
| Premature delivery 10036595 PT |
| Premature labour 10036600 PT |
| Premature rupture of membranes 10036603 PT |
| Premature separation of placenta 10036608 PT |
| Prenatal screening test abnormal 10069151 PT |
| Preterm premature rupture of membranes 10073024 PT |


## 18.2 Adverse Events Related to Pregnancy

Events pertaining to PTs from MedDRA SMQ "Pregnancy and neonatal topics" with rationales for exclusion in the AEs related to pregnancy.

| Unique<br>Subject<br>Identifie | Reported Term for the Clinical Event | Analysis<br>Preferred<br>Term<br>Code | Analysis<br>Preferred Term | Start<br>Date/Time<br>of Clinical<br>Event | End<br>Date/Time<br>of<br>Adverse<br>Event | Severity/Intensity | Causality | Outcome of<br>Event | Relations<br>hip to<br>Non-<br>Study<br>Treatment | Action Taken with<br>Study Treatment | Serious<br>Event | AE<br>related to<br>pregancy<br>? | Reason for exclusion |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| PPD | | | | | | | | | | | | | |















| 18.3 | <b>AESI: Opportunistic Infections</b> |
|------|---------------------------------------|


## 18.4 AESI Herpes Zoster


# 18.5 Malignant or Unspecified Tumours (SMQ 20000091)


| Name Code Level |
|---------------------------------------------------------------------|
| Naurius I - aug I usau Is aug aug un fun at aug |
| Marginal zone lymphoma refractory 10077534 PT |
| Marginal zone lymphoma stage I 10077529 PT |
| Marginal zone lymphoma stage II 10077530 PT |
| Marginal zone lymphoma stage III 10077531 PT |
| Marginal zone lymphoma stage IV 10077532 PT |
| Mastocytic leukaemia 10056450 PT |
| Mature B-cell type acute leukaemia 10026945 PT |
| Metastases to bone marrow 10051662 PT |
| Metastases to lymph nodes 10027459 PT |
| Metastases to spleen 10051682 PT |
| Metastatic lymphoma 10071541 PT |
| Minimal residual disease 10079987 PT |
| Monocytic leukaemia in remission 10061295 PT |
| Mycosis fungoides 10028483 PT |
| Mycosis fungoides recurrent 10028501 PT |
| Mycosis fungoides refractory 10028502 PT |
| Mycosis fungoides stage I 10028503 PT |
| Mycosis fungoides stage II 10028504 PT |
| Mycosis fungoides stage III 10028505 PT |
| Mycosis fungoides stage IV 10028506 PT |
| Myeloblastoma 10051141 PT |
| Myeloid leukaemia 10028549 PT |
| Myeloid leukaemia in remission 10061301 PT |
| Natural killer-cell leukaemia 10028811 PT |
| Natural killer-cell lymphoblastic lymphoma 10058975 PT |
| Neonatal leukaemia 10028958 PT |
| Nodal marginal zone B-cell lymphoma 10029460 PT |
| Nodal marginal zone B-cell lymphoma recurrent 10029463 PT |
| Nodal marginal zone B-cell lymphoma refractory 10029464 PT |
| Nodal marginal zone B-cell lymphoma stage I 10029465 PT |
| Nodal marginal zone B-cell lymphoma stage II 10029466 PT |
| Nodal marginal zone B-cell lymphoma stage III 10029467 PT |
| Nodal marginal zone B-cell lymphoma stage IV 10029468 PT |
| Nodular lymphocyte predominant Hodgkin lymphoma 10080201 PT |
| Non-Hodgkin's lymphoma 10029547 PT |
| Non-Hodgkin's lymphoma metastatic 10071535 PT |
| Non-Hodgkin's lymphoma stage I 10029602 PT |
| Non-Hodgkin's lymphoma stage II 10029603 PT |
| Non-Hodgkin's lymphoma stage III 10029604 PT |
| Non-Hodgkin's lymphoma stage IV 10029605 PT |
| Non-Hodgkin's lymphoma transformed recurrent 10061871 PT |
| Non-Hodgkin's lymphoma unspecified histology aggressive 10063908 PT |


| NameCodeLevelAcral lentiginous melanoma10000583PTAcral lentiginous melanoma stage I10000585PTAcral lentiginous melanoma stage II10000586PTAcral lentiginous melanoma stage III10000587PTAcral lentiginous melanoma stage IV10000588PTAdenocarcinoma10001141PT |
|---|
| Acral lentiginous melanoma stage I 10000585 PT Acral lentiginous melanoma stage II 10000586 PT Acral lentiginous melanoma stage III 10000587 PT Acral lentiginous melanoma stage IV 10000588 PT |
| Acral lentiginous melanoma stage II 10000586 PT Acral lentiginous melanoma stage III 10000587 PT Acral lentiginous melanoma stage IV 10000588 PT |
| Acral lentiginous melanoma stage III 10000587 PT Acral lentiginous melanoma stage IV 10000588 PT |
| Acral lentiginous melanoma stage IV 10000588 PT |
| Adenocarcinoma 10001141 PT |
| Adenocarcinoma gastric 10001150 PT |
| Adenocarcinoma of appendix 10073359 PT |
| Adenocarcinoma of colon 10001167 PT |
| Adenocarcinoma of salivary gland 10068068 PT |
| Adenocarcinoma of the cervix 10001197 PT |
| Adenocarcinoma pancreas 10052747 PT |
| Adenoid cystic carcinoma 10053231 PT |
| Adenoid cystic carcinoma of external auditory canal 10078057 PT |
| Adenoid cystic carcinoma of salivary gland 10073370 PT |
| Adenosquamous carcinoma of the cervix 10001244 PT |
| Adenosquamous carcinoma of vagina 10073978 PT |
| Adenosquamous cell carcinoma 10068873 PT |
| Adenosquamous cell lung cancer 10001245 PT |
| Adenosquamous cell lung cancer recurrent 10001247 PT |
| Adenosquamous cell lung cancer stage 0 10001248 PT |
| Adenosquamous cell lung cancer stage I 10001249 PT |
| Adenosquamous cell lung cancer stage II 10001250 PT |
| Adenosquamous cell lung cancer stage III 10001251 PT |
| Adenosquamous cell lung cancer stage IV 10001254 PT |
| Adrenal gland cancer 10073152 PT |
| Adrenal gland cancer metastatic 10055095 PT |
| Adrenocortical carcinoma 10001388 PT |
| Aesthesioneuroblastoma 10001433 PT |
| Alveolar rhabdomyosarcoma 10065867 PT |
| Alveolar soft part sarcoma 10001882 PT |
| Alveolar soft part sarcoma metastatic 10001884 PT |
| Alveolar soft part sarcoma recurrent 10001887 PT |
| Anal cancer 10061424 PT |
| Anal cancer metastatic 10055096 PT |
| Anal cancer recurrent 10002133 PT |
| Anal cancer stage 0 10002134 PT |
| Anal cancer stage I 10002135 PT |
| Anal cancer stage II 10002136 PT |
| Anal cancer stage III 10002137 PT |
| Anal cancer stage IV 10002138 PT |
| Anal squamous cell carcinoma 10073358 PT |
| Anaplastic astrocytoma 10002224 PT |
| Anaplastic meningioma 10073127 PT |


| Name Code Level Colon cancer stage 0 10063523 PT Colon cancer stage 1 10009953 PT Colon cancer stage III 10009954 PT Colon cancer stage IVI 10009955 PT Color cancer stage IV 10009956 PT Colorectal adenocarcinoma 10052360 PT Colorectal cancer 10061451 PT Colorectal cancer metastatic 10052358 PT Colorectal cancer recurrent 10010030 PT Colorectal cancer stage I 10010033 PT Colorectal cancer stage III 10010033 PT Colorectal cancer stage IV 10010034 PT Colorectal carcinoma stage 0 10010038 PT Congenital fibrosarcoma 10065859 PT Congenital malignant neoplasm 10073470 PT Conjunctival melanoma 1006384 PT Cystadenocarcinoma ovary 10054912 PT Cystadenocarcinoma pancreas 10065908 PT Dedifferenti |
|---|
| Colon cancer stage I Colon cancer stage II Colon cancer stage III Colon cancer stage III Colon cancer stage III Colon cancer stage IV Colon cancer stage IV Colorectal adenocarcinoma 10052360 Colorectal cancer 10061451 Colorectal cancer metastatic 10052358 Colorectal cancer recurrent 10010030 Colorectal cancer stage I Colorectal cancer stage I 10010032 Colorectal cancer stage I 10010033 Colorectal cancer stage II Colorectal cancer stage II 10010034 Colorectal cancer stage II Colorectal cancer stage IV Colorectal carcinoma stage 0 10010038 Congenital fibrosarcoma 10065859 Congenital malignant neoplasm 10073492 Congenital malignant neoplasm 10073492 Conjunctival melanoma 10066384 Cystadenocarcinoma ovary 10054912 Cystadenocarcinoma pancreas 10065908 Cystadenocarcinoma pancreas 10065908 Cystadenocarcinoma protuberans Dermatofibrosarcoma protuberans metastatic 10073574 Colorectal cancer stage IV Colorectal cancer stage II Colorect |
| Colon cancer stage II 10009954 PT Colon cancer stage III 10009955 PT Colon cancer stage IV 10009956 PT Colorectal adenocarcinoma 10052360 PT Colorectal cancer 10061451 PT Colorectal cancer metastatic 10052358 PT Colorectal cancer recurrent 10010030 PT Colorectal cancer stage I 10010032 PT Colorectal cancer stage III 10010033 PT Colorectal cancer stage IV 10010034 PT Colorectal carcinoma stage 0 10010035 PT Congenital fibrosarcoma 10065859 PT Congenital malignant neoplasm 10073492 PT Congenital retinoblastoma 10073470 PT Conjunctival melanoma 10066384 PT Cystadenocarcinoma ovary 10054912 PT Cystadenocarcinoma pancreas 10065908 PT Dedifferentiated liposarcoma 10073135 PT Dermatofibrosarcoma protuberans 10057070 PT |
| Colon cancer stage III 10009955 PT Colon cancer stage IV 10009956 PT Colorectal adenocarcinoma 10052360 PT Colorectal cancer 10061451 PT Colorectal cancer metastatic 10052358 PT Colorectal cancer recurrent 10010030 PT Colorectal cancer stage I 10010032 PT Colorectal cancer stage II 10010033 PT Colorectal cancer stage III 10010034 PT Colorectal cancer stage III 10010035 PT Colorectal cancer stage IV 10010035 PT Colorectal cancer stage IV 10010038 PT Congenital fibrosarcoma 10065859 PT Congenital malignant neoplasm 10073492 PT Congenital retinoblastoma 10073470 PT Conjunctival melanoma 10066384 PT Cystadenocarcinoma ovary 10054912 PT Cystadenocarcinoma pancreas 10065908 PT Dedifferentiated liposarcoma 10073135 PT Dermatofibrosarcoma protuberans metastatic 10073574 PT |
| Colon cancer stage IV Colorectal adenocarcinoma 10052360 PT Colorectal cancer 10061451 PT Colorectal cancer metastatic 10052358 PT Colorectal cancer recurrent 10010030 PT Colorectal cancer stage I 10010032 PT Colorectal cancer stage II 10010033 PT Colorectal cancer stage III 10010034 PT Colorectal cancer stage III 10010035 PT Colorectal cancer stage IV 10010035 PT Colorectal cancer stage IV 10010036 PT Colorectal cancer stage IV 10010037 PT Colorectal cancer stage IV Congenital fibrosarcoma 10065859 PT Congenital malignant neoplasm 10073492 PT Congenital retinoblastoma 10073470 PT Conjunctival melanoma 10066384 PT Cystadenocarcinoma ovary 10054912 PT Cystadenocarcinoma pancreas 10065908 PT Dedifferentiated liposarcoma 10073135 PT Dermatofibrosarcoma protuberans metastatic |
| Colorectal adenocarcinoma Colorectal cancer Colorectal cancer etastatic Colorectal cancer metastatic Colorectal cancer recurrent Colorectal cancer stage I Colorectal cancer stage II Colorectal cancer stage III Colorectal cancer stage III Colorectal cancer stage IV Colorectal cancer stage IV Colorectal carcinoma stage 0 Congenital fibrosarcoma Congenital malignant neoplasm Congenital retinoblastoma Conjunctival melanoma Cystadenocarcinoma ovary Cystadenocarcinoma pancreas Dedifferentiated liposarcoma Dermatofibrosarcoma protuberans metastatic 10052350 PT Colorectal cancer stage IV 10010032 PT Colorectal cancer stage IV 10010035 PT Colorectal carcinoma stage 0 10010038 PT Conjunctival melanoma 10065859 PT Congenital retinoblastoma 10073470 PT Cystadenocarcinoma ovary 10054912 PT Cystadenocarcinoma pancreas 10065908 PT Dermatofibrosarcoma protuberans metastatic |
| Colorectal cancer Colorectal cancer metastatic 10052358 PT Colorectal cancer recurrent 10010030 PT Colorectal cancer stage I 10010032 PT Colorectal cancer stage II 10010033 PT Colorectal cancer stage III 10010033 PT Colorectal cancer stage III 10010034 PT Colorectal cancer stage IV 10010035 PT Colorectal cancer stage IV 10010035 PT Colorectal carcinoma stage O 10010038 PT Congenital fibrosarcoma 10065859 PT Congenital malignant neoplasm 10073492 PT Congenital retinoblastoma 10073470 PT Conjunctival melanoma 10066384 PT Cystadenocarcinoma ovary 10054912 PT Cystadenocarcinoma pancreas 10065908 PT Dedifferentiated liposarcoma 10073135 PT Dermatofibrosarcoma protuberans metastatic 10073574 PT |
| Colorectal cancer metastatic Colorectal cancer recurrent Colorectal cancer stage I Colorectal cancer stage I Colorectal cancer stage II Colorectal cancer stage III Colorectal cancer stage III Colorectal cancer stage IV Colorectal carcinoma stage O Congenital fibrosarcoma Congenital malignant neoplasm Congenital retinoblastoma Conjunctival melanoma Cystadenocarcinoma ovary Cystadenocarcinoma pancreas Dedifferentiated liposarcoma Dermatofibrosarcoma protuberans 10052358 PT 10010030 PT 10010033 PT 10010035 PT 10010038 PT 10065859 PT Congenital retinoblastoma 10073470 PT Cystadenocarcinoma ovary 10054912 PT Cystadenocarcinoma pancreas 10065908 PT Dermatofibrosarcoma protuberans 10057070 PT Dermatofibrosarcoma protuberans metastatic |
| Colorectal cancer recurrent10010030PTColorectal cancer stage I10010032PTColorectal cancer stage III10010033PTColorectal cancer stage IV10010035PTColorectal carcinoma stage 010010038PTCongenital fibrosarcoma10065859PTCongenital malignant neoplasm10073492PTCongenital retinoblastoma10073470PTConjunctival melanoma10066384PTCystadenocarcinoma ovary10054912PTCystadenocarcinoma pancreas10073135PTDedifferentiated liposarcoma10073135PTDermatofibrosarcoma protuberans10057070PTDermatofibrosarcoma protuberans metastatic10073574PT |
| Colorectal cancer stage I Colorectal cancer stage II Colorectal cancer stage III Colorectal cancer stage III Colorectal cancer stage IV Colorectal carcinoma stage 0 Colorectal carcinoma stage 0 Congenital fibrosarcoma Congenital malignant neoplasm Congenital retinoblastoma Conjunctival melanoma Conjunctival melanoma Cystadenocarcinoma ovary Cystadenocarcinoma pancreas Dedifferentiated liposarcoma Dermatofibrosarcoma protuberans Dermatofibrosarcoma protuberans metastatic 10010032 PT 10010033 PT 10010035 PT 10073470 PT 10054912 PT 10057070 PT 10057070 PT |
| Colorectal cancer stage III Colorectal cancer stage IIII Colorectal cancer stage IV Colorectal cancer stage IV Colorectal carcinoma stage 0 Congenital fibrosarcoma Congenital malignant neoplasm Congenital retinoblastoma Conjunctival melanoma Conjunctival melanoma Cystadenocarcinoma ovary Cystadenocarcinoma pancreas Dedifferentiated liposarcoma Dermatofibrosarcoma protuberans metastatic 10010033 PT 10010035 PT 10010035 PT 10010038 PT 10065859 PT 10073470 PT 10066384 PT 10065908 PT 10073135 PT 10073135 PT |
| Colorectal cancer stage III Colorectal cancer stage IV Colorectal carcinoma stage 0 Congenital fibrosarcoma Congenital malignant neoplasm Congenital retinoblastoma Conjunctival melanoma Cystadenocarcinoma ovary Cystadenocarcinoma pancreas Dedifferentiated liposarcoma Dermatofibrosarcoma protuberans Dermatofibrosarcoma protuberans metastatic 10010034 PT 10010038 PT 10065859 PT 10073492 PT 10073470 PT 10054912 PT 10054912 PT 10057070 PT 10057070 PT |
| Colorectal cancer stage IV Colorectal carcinoma stage 0 10010038 PT Congenital fibrosarcoma 10065859 PT Congenital malignant neoplasm 10073492 PT Congenital retinoblastoma 10073470 PT Conjunctival melanoma 10066384 PT Cystadenocarcinoma ovary 10054912 PT Cystadenocarcinoma pancreas 10065908 PT Dedifferentiated liposarcoma 10073135 PT Dermatofibrosarcoma protuberans 10057070 PT |
| Colorectal carcinoma stage 0 Congenital fibrosarcoma 10065859 PT Congenital malignant neoplasm 10073492 PT Congenital retinoblastoma 10073470 PT Conjunctival melanoma 10066384 PT Cystadenocarcinoma ovary 10054912 PT Cystadenocarcinoma pancreas 10065908 PT Dedifferentiated liposarcoma 10073135 PT Dermatofibrosarcoma protuberans 10057070 PT Dermatofibrosarcoma protuberans metastatic |
| Congenital fibrosarcoma10065859PTCongenital malignant neoplasm10073492PTCongenital retinoblastoma10073470PTConjunctival melanoma10066384PTCystadenocarcinoma ovary10054912PTCystadenocarcinoma pancreas10065908PTDedifferentiated liposarcoma10073135PTDermatofibrosarcoma protuberans10057070PTDermatofibrosarcoma protuberans metastatic10073574PT |
| Congenital malignant neoplasm10073492PTCongenital retinoblastoma10073470PTConjunctival melanoma10066384PTCystadenocarcinoma ovary10054912PTCystadenocarcinoma pancreas10065908PTDedifferentiated liposarcoma10073135PTDermatofibrosarcoma protuberans10057070PTDermatofibrosarcoma protuberans metastatic10073574PT |
| Congenital retinoblastoma10073470PTConjunctival melanoma10066384PTCystadenocarcinoma ovary10054912PTCystadenocarcinoma pancreas10065908PTDedifferentiated liposarcoma10073135PTDermatofibrosarcoma protuberans10057070PTDermatofibrosarcoma protuberans metastatic10073574PT |
| Conjunctival melanoma10066384PTCystadenocarcinoma ovary10054912PTCystadenocarcinoma pancreas10065908PTDedifferentiated liposarcoma10073135PTDermatofibrosarcoma protuberans10057070PTDermatofibrosarcoma protuberans metastatic10073574PT |
| Cystadenocarcinoma ovary10054912PTCystadenocarcinoma pancreas10065908PTDedifferentiated liposarcoma10073135PTDermatofibrosarcoma protuberans10057070PTDermatofibrosarcoma protuberans metastatic10073574PT |
| Cystadenocarcinoma pancreas10065908PTDedifferentiated liposarcoma10073135PTDermatofibrosarcoma protuberans10057070PTDermatofibrosarcoma protuberans metastatic10073574PT |
| Dedifferentiated liposarcoma10073135PTDermatofibrosarcoma protuberans10057070PTDermatofibrosarcoma protuberans metastatic10073574PT |
| Dermatofibrosarcoma protuberans metastatic 10073574 PT |
| · |
| Desmoplastic melanoma 10072449 PT |
| Desmoplastic mesothelioma 10073063 PT |
| Desmoplastic small round cell tumour 10064581 PT |
| Ductal adenocarcinoma of pancreas 10073364 PT |
| Ear neoplasm malignant 10055017 PT |
| Eccrine carcinoma 10069680 PT |
| Embryonal rhabdomyosarcoma 10065868 PT |
| Endocrine neoplasm malignant 10061122 PT |
| Endometrial adenocarcinoma 10014720 PT |
| Endometrial cancer 10014733 PT |
| Endometrial cancer metastatic 10014734 PT |
| Endometrial cancer recurrent 10014736 PT |
| Endometrial cancer stage 0 10014737 PT |
| Endometrial cancer stage I 10014738 PT |
| Endometrial cancer stage II 10014739 PT |
| Endometrial cancer stage III 10014740 PT |
| Endometrial cancer stage IV 10014741 PT |
| Endometrial sarcoma 10057649 PT |
| Endometrial sarcoma metastatic 10067065 PT |
| Endometrial sarcoma recurrent 10067064 PT |
| Endometrial stromal sarcoma 10048397 PT |


| Name Code Level Fallopian tube cancer stage IV 10016187 PT Familial medullary thyroid cancer 10073153 PT Female reproductive tract carcinoma in situ 10061154 PT Fibrosarcoma 10016632 PT Fibrosarcoma metastatic 10016935 PT Follicular thyroid cancer 10016935 PT Gallbladder adenocarcinoma 10016935 PT Gallbladder adenosquamous carcinoma 10073067 PT Gallbladder adenosquamous carcinoma 10073067 PT Gallbladder cancer 10017614 PT Gallbladder cancer extage il 10017614 PT Gallbladder cancer stage 0 10059316 PT Gallbladder cancer stage 1 10059317 PT Gallbladder cancer stage II 10058281 PT Gallbladder cancer stage II 10058282 PT Gallbladder squamous cell carcinoma 1007308 PT Gallbladder squamous cell carcinoma 10017708 PT Gastric cancer 10017708 |
|---|
| Familial medullary thyroid cancer 10073153 PT Female reproductive tract carcinoma in situ 10061154 PT Fibrosarcoma 10016632 PT Fibrosarcoma metastatic 10016635 PT Follicular thyroid cancer 10016935 PT Gallbladder adenocarcinoma 10073067 PT Gallbladder adenosquamous carcinoma 10073067 PT Gallbladder cancer 10017614 PT Gallbladder cancer metastatic 1006879 PT Gallbladder cancer stage 0 10059316 PT Gallbladder cancer stage I 10059316 PT Gallbladder cancer stage II 10058281 PT Gallbladder cancer stage III 10058282 PT Gallbladder squamous cell carcinoma 10073068 PT Ganglioglioma 10017701 PT Gastric cancer stage II 10017708 PT Gastric cancer stage I 10017768 PT Gastric cancer stage I 10017769 PT Gastric cancer stage II 10017769 < |
| Female reproductive tract carcinoma in situ Fibrosarcoma 10016632 PT Fibrosarcoma 10016632 Fibrosarcoma metastatic 10016635 FT Follicular thyroid cancer 1001635 FT Gallbladder adenocarcinoma 10078067 Gallbladder adenosquamous carcinoma 10073067 FT Gallbladder cancer 10017614 FT Gallbladder cancer metastatic 10066879 Gallbladder cancer recurrent 10017619 FT Gallbladder cancer stage 0 10059316 FT Gallbladder cancer stage 1 10059316 FT Gallbladder cancer stage 1 10059316 FT Gallbladder cancer stage II Gallbladder cancer stage III 10058281 FT Gallbladder cancer stage III Gallbladder squamous cell carcinoma 10073068 FT Ganglionglioma 10017701 FT Ganglioneuroblastoma 10017708 FT Gastric cancer 10017758 FT Gastric cancer stage I G |
| Fibrosarcoma 10016632 PT Fibrosarcoma metastatic 10016635 PT Follicular thyroid cancer 10016935 PT Gallbladder adenocarcinoma 10058286 PT Gallbladder adenosquamous carcinoma 10073067 PT Gallbladder cancer 10017614 PT Gallbladder cancer metastatic 10066879 PT Gallbladder cancer stage 0 10017619 PT Gallbladder cancer stage 1 10059316 PT Gallbladder cancer stage 8 10059317 PT Gallbladder cancer stage 9 10059317 PT Gallbladder cancer stage 11 10058281 PT Gallbladder cancer stage 18 10058282 PT Gallbladder squamous cell carcinoma 10078382 PT Gallbladder squamous cell carcinoma 10017701 PT Ganglioglioma 10017701 PT Gastric cancer 10017708 PT Gastric cancer stage 0 10017762 PT Gastric cancer stage 1 10017763 PT |
| Fibrosarcoma metastatic Follicular thyroid cancer Follicular thyroid cancer Gallbladder adenocarcinoma Gallbladder adenosquamous carcinoma Gallbladder cancer Gallbladder cancer Gallbladder cancer metastatic Gallbladder cancer metastatic Gallbladder cancer recurrent Gallbladder cancer stage 0 Gallbladder cancer stage I Gallbladder cancer stage II Gallbladder squamous cell carcinoma 10073068 PT Ganglioglioma 10017701 PT Ganglioneuroblastoma 10017708 PT Gastric cancer 10017758 PT Gastric cancer recurrent 10017762 PT Gastric cancer stage I 10017763 PT Gastric cancer stage II 10017764 PT Gastric cancer stage II 10017765 PT Gastric cancer stage II 10017765 PT Gastric cancer stage II 10017765 PT Gastric sarcoma 10055008 PT Gastrionam malignant 10051709 PT Gastrointestinal adenocarcinoma 10081003 PT |
| Follicular thyroid cancer Gallbladder adenocarcinoma Gallbladder adenosquamous carcinoma Gallbladder cancer Gallbladder cancer Gallbladder cancer metastatic Gallbladder cancer metastatic Gallbladder cancer recurrent Gallbladder cancer stage 0 Gallbladder cancer stage 1 Ganglionma 10017701 FT Gastric cancer Ganglioneuroblastoma 10017702 FT Gastric cancer stage 0 10017762 FT Gastric cancer stage 1 10017763 FT Gastric cancer stage 1 10017764 FT Gastric cancer stage 1 10017765 FT Gastric cancer stage 1 10017761 FT Gastric cancer stage 1 10017761 FT Gastric cancer stage 1 10017761 FT Ga |
| Gallbladder adenocarcinoma Gallbladder adenosquamous carcinoma Gallbladder cancer Gallbladder cancer Gallbladder cancer metastatic Gallbladder cancer metastatic Gallbladder cancer recurrent Gallbladder cancer stage 0 Gallbladder cancer stage 1 Ganglioglioma 10017701 PT Ganglioglioma 10017702 PT Gastric cancer 10017758 PT Gastric cancer stage 0 10017762 PT Gastric cancer stage 1 10017763 PT Gastric cancer stage 1 10017764 PT Gastric cancer stage 1 10017765 PT Gastric cancer stage 1 10017769 PT Gastric cancer stage 1 10017769 PT Gastric cancer stage 1 10051709 PT Gastric sarcoma 10051709 PT Gastrionma malignant 10051709 PT Gastrointestinal adenocarcinoma 10081003 PT Gastrointestinal cancer metastatic |
| Gallbladder adenosquamous carcinoma Gallbladder cancer Gallbladder cancer metastatic Gallbladder cancer metastatic 10066879 FT Gallbladder cancer recurrent 10017619 FT Gallbladder cancer stage 0 10059316 FT Gallbladder cancer stage I Gallbladder cancer stage II Gallbladder cancer stage II Gallbladder cancer stage III Gallbladder squamous cell carcinoma 10073068 FT Ganglioneuroblastoma 10017701 FT Ganglioneuroblastoma 10017708 FT Gastric cancer 10017758 FT Gastric cancer recurrent 10017762 FT Gastric cancer stage 0 10017763 FT Gastric cancer stage I 10017764 FT Gastric cancer stage II 10017765 FT Gastric cancer stage II 10017767 FT Gastric cancer stage II 10017769 FT Gastric cancer stage II 10055008 FT Gastrionam malignant 10051709 FT Gastrointestinal adenocarcinoma 10081003 FT Gastrointestinal cancer metastatic |
| Gallbladder cancer10017614PTGallbladder cancer metastatic10066879PTGallbladder cancer recurrent10017619PTGallbladder cancer stage 010059316PTGallbladder cancer stage I10059317PTGallbladder cancer stage III10058281PTGallbladder cancer stage IVI10058282PTGallbladder squamous cell carcinoma10073068PTGanglioglioma10017701PTGastric cancer10017768PTGastric cancer recurrent10017761PTGastric cancer stage I10017762PTGastric cancer stage I10017763PTGastric cancer stage I10017765PTGastric cancer stage III10017765PTGastric cancer stage III10017765PTGastric cancer stage IV10061967PTGastric cancer stage IV10061967PTGastric man malignant10055008PTGastroenteropancreatic neuroendocrine tumour disease10077559PTGastrointestinal adenocarcinoma10081003PTGastrointestinal cancer metastatic10053548PT |
| Gallbladder cancer metastatic Gallbladder cancer recurrent Gallbladder cancer recurrent Gallbladder cancer stage 0 10059316 PT Gallbladder cancer stage 1 10059317 PT Gallbladder cancer stage II Gallbladder cancer stage III Gallbladder cancer stage III Gallbladder cancer stage III Gallbladder cancer stage III Gallbladder cancer stage III Gallbladder cancer stage IV Gallbladder squamous cell carcinoma 10058283 Gallbladder squamous cell carcinoma 10073068 Ganglioglioma 10017701 PT Ganglioneuroblastoma 10017708 PT Gastric cancer 10017758 PT Gastric cancer recurrent 10017761 PT Gastric cancer stage 0 10017762 PT Gastric cancer stage I 10017763 PT Gastric cancer stage II 10017765 PT Gastric cancer stage III 10017765 PT Gastric cancer stage IV 10061967 PT Gastric sarcoma 10055008 PT Gastrionam malignant 10051709 PT Gastroenteropancreatic neuroendocrine tumour disease 10077559 PT Gastrointestinal adenocarcinoma 10081003 PT Gastrointestinal cancer metastatic |
| Gallbladder cancer recurrent Gallbladder cancer stage 0 10059316 PT Gallbladder cancer stage 1 10059317 PT Gallbladder cancer stage II Gallbladder cancer stage III Gallbladder cancer stage III Gallbladder cancer stage III Gallbladder cancer stage III Gallbladder cancer stage IV Gallbladder squamous cell carcinoma 10058283 PT Gallbladder squamous cell carcinoma 10073068 PT Ganglioneuroblastoma 10017701 PT Ganglioneuroblastoma 10017708 PT Gastric cancer 10017758 PT Gastric cancer recurrent 10017761 PT Gastric cancer stage 0 10017762 PT Gastric cancer stage I 10017763 PT Gastric cancer stage II 10017764 PT Gastric cancer stage III 10017765 PT Gastric cancer stage III 10017765 PT Gastric cancer stage IV 10061967 PT Gastric sarcoma 10055008 PT Gastrionam malignant 10051709 PT Gastroenteropancreatic neuroendocrine tumour disease 10077559 PT Gastrointestinal adenocarcinoma 10081003 PT Gastrointestinal cancer metastatic |
| Gallbladder cancer stage I Gallbladder cancer stage I Gallbladder cancer stage II Gallbladder cancer stage III Gallbladder cancer stage III Gallbladder cancer stage III Gallbladder cancer stage IV Gallbladder squamous cell carcinoma Ganglioglioma 10017701 FT Ganglioneuroblastoma 10017708 FT Gastric cancer 10017758 FT Gastric cancer recurrent 10017761 FT Gastric cancer stage I Gastric cancer stage I Gastric cancer stage I Gastric cancer stage I Gastric cancer stage II Gastric cancer stage II Gastric cancer stage II Gastric cancer stage IV Gastric cancer stage IV Gastric cancer stage IV Gastric cancer stage II Gastric cancer stage IV Gastric cancer stage IV Gastric sarcoma 10017765 FT Gastric sarcoma 10051709 FT Gastrioma malignant Gastroenteropancreatic neuroendocrine tumour disease 10077559 FT Gastrointestinal adenocarcinoma 10081003 FT Gastrointestinal cancer metastatic |
| Gallbladder cancer stage I Gallbladder cancer stage II Gallbladder cancer stage III Gallbladder cancer stage III Gallbladder cancer stage IV Gallbladder cancer stage IV Gallbladder squamous cell carcinoma 10073068 PT Ganglioneuroblastoma 10017701 PT Ganglioneuroblastoma 10017708 PT Gastric cancer 10017758 PT Gastric cancer recurrent 10017761 PT Gastric cancer stage 0 10017762 PT Gastric cancer stage I 10017763 PT Gastric cancer stage II 10017764 PT Gastric cancer stage II 10017765 PT Gastric cancer stage IV 10017765 PT Gastric cancer stage IV 10061967 PT Gastric sarcoma 10055008 PT Gastrionam malignant 10051709 PT Gastroenteropancreatic neuroendocrine tumour disease 10077559 PT Gastrointestinal adenocarcinoma 10081003 PT Gastrointestinal cancer metastatic |
| Gallbladder cancer stage II Gallbladder cancer stage III Gallbladder cancer stage IV Gallbladder cancer stage IV Gallbladder squamous cell carcinoma Ganglioglioma Ganglioneuroblastoma Gastric cancer Gastric cancer recurrent Gastric cancer stage I Gastric cancer stage II Gastric cancer stage II Gastric cancer stage II Gastric cancer stage IV Gastric sarcoma Gastrinoma malignant Gastrointestinal adenocarcinoma 10081003 PT Gastrointestinal cancer metastatic |
| Gallbladder cancer stage III Gallbladder cancer stage IV Gallbladder squamous cell carcinoma Ganglioglioma 10073068 FT Ganglioneuroblastoma 10017701 FT Gastric cancer 10017758 Gastric cancer recurrent 10017761 FT Gastric cancer stage 0 10017762 FT Gastric cancer stage I 10017763 FT Gastric cancer stage II 10017764 FT Gastric cancer stage II 10017765 FT Gastric cancer stage III 10017765 FT Gastric cancer stage III 10017765 FT Gastric cancer stage III 10017765 FT Gastric cancer stage II 10017765 FT Gastric sarcoma 10055008 FT Gastrioma malignant 10051709 FT Gastroenteropancreatic neuroendocrine tumour disease 10077559 FT Gastrointestinal adenocarcinoma 10081003 FT Gastrointestinal cancer metastatic |
| Gallbladder cancer stage IV Gallbladder squamous cell carcinoma Ganglioglioma 10073068 PT Ganglioneuroblastoma 10017701 PT Gastric cancer 10017758 Gastric cancer recurrent 10017761 PT Gastric cancer stage 0 10017762 PT Gastric cancer stage II 10017763 PT Gastric cancer stage III 10017765 PT Gastric cancer stage IV 10017765 PT Gastric cancer stage IV 10061967 Gastric cancer stage IV Gastric cancer stage IV Gastric cancer stage IV Gastric cancer stage IV Gastric cancer stage IV Gastric sarcoma 10055008 Gastrioma malignant 10051709 PT Gastroenteropancreatic neuroendocrine tumour disease 10077559 PT Gastrointestinal adenocarcinoma 10081003 PT Gastrointestinal cancer metastatic |
| Gallbladder squamous cell carcinoma10073068PTGanglioglioma10017701PTGanglioneuroblastoma10017708PTGastric cancer10017758PTGastric cancer recurrent10017761PTGastric cancer stage 010017762PTGastric cancer stage I10017763PTGastric cancer stage III10017764PTGastric cancer stage IVI10061967PTGastric sarcoma10055008PTGastrinoma malignant10051709PTGastroenteropancreatic neuroendocrine tumour disease10077559PTGastrointestinal adenocarcinoma10081003PTGastrointestinal cancer metastatic10053548PT |
| Ganglioglioma10017701PTGanglioneuroblastoma10017708PTGastric cancer10017758PTGastric cancer recurrent10017761PTGastric cancer stage 010017762PTGastric cancer stage I10017763PTGastric cancer stage III10017764PTGastric cancer stage IVI10061967PTGastric sarcoma10055008PTGastrinoma malignant10051709PTGastroenteropancreatic neuroendocrine tumour disease10077559PTGastrointestinal adenocarcinoma10081003PTGastrointestinal cancer metastatic10053548PT |
| Ganglioneuroblastoma10017708PTGastric cancer10017758PTGastric cancer recurrent10017761PTGastric cancer stage 010017762PTGastric cancer stage I10017763PTGastric cancer stage III10017764PTGastric cancer stage IVI10017765PTGastric sarcoma10055008PTGastrinoma malignant10051709PTGastroenteropancreatic neuroendocrine tumour disease10077559PTGastrointestinal adenocarcinoma10081003PTGastrointestinal cancer metastatic10053548PT |
| Gastric cancer10017758PTGastric cancer recurrent10017761PTGastric cancer stage 010017762PTGastric cancer stage I10017763PTGastric cancer stage III10017764PTGastric cancer stage IVI10017765PTGastric sarcoma10055008PTGastrinoma malignant10051709PTGastroenteropancreatic neuroendocrine tumour disease10077559PTGastrointestinal adenocarcinoma10081003PTGastrointestinal cancer metastatic10053548PT |
| Gastric cancer recurrent Gastric cancer stage 0 10017762 PT Gastric cancer stage I 10017763 PT Gastric cancer stage II 10017764 PT Gastric cancer stage III 10017765 Gastric cancer stage IV 10061967 PT Gastric sarcoma 10055008 Gastrinoma malignant 10051709 PT Gastroenteropancreatic neuroendocrine tumour disease 10077559 PT Gastrointestinal adenocarcinoma 10081003 PT Gastrointestinal cancer metastatic |
| Gastric cancer stage 0 Gastric cancer stage I Gastric cancer stage II Gastric cancer stage III Gastric cancer stage III Gastric cancer stage IV Gastric cancer stage IV Gastric sarcoma Gastric sarcoma Gastrinoma malignant Gastroenteropancreatic neuroendocrine tumour disease Gastrointestinal adenocarcinoma Gastrointestinal cancer metastatic 10017762 PT 10017763 PT 10017765 PT 10051709 PT 10081003 PT 10081003 PT |
| Gastric cancer stage I 10017763 PT Gastric cancer stage II 10017764 PT Gastric cancer stage III 10017765 PT Gastric cancer stage IV 10061967 PT Gastric sarcoma 10055008 PT Gastrinoma malignant 10051709 PT Gastroenteropancreatic neuroendocrine tumour disease 10077559 PT Gastrointestinal adenocarcinoma 10081003 PT Gastrointestinal cancer metastatic 10053548 PT |
| Gastric cancer stage II 10017764 PT Gastric cancer stage III 10017765 PT Gastric cancer stage IV 10061967 PT Gastric sarcoma 10055008 PT Gastrinoma malignant 10051709 PT Gastroenteropancreatic neuroendocrine tumour disease 10077559 PT Gastrointestinal adenocarcinoma 10081003 PT Gastrointestinal cancer metastatic 10053548 PT |
| Gastric cancer stage III Gastric cancer stage IV Gastric sarcoma 10061967 PT Gastric sarcoma 10055008 Gastrinoma malignant 10051709 FT Gastroenteropancreatic neuroendocrine tumour disease 10077559 FT Gastrointestinal adenocarcinoma 10081003 FT Gastrointestinal cancer metastatic 10053548 FT |
| Gastric cancer stage IV Gastric sarcoma 10061967 PT Gastric sarcoma 10055008 PT Gastrinoma malignant 10051709 PT Gastroenteropancreatic neuroendocrine tumour disease 10077559 PT Gastrointestinal adenocarcinoma 10081003 PT Gastrointestinal cancer metastatic 10053548 PT |
| Gastric sarcoma10055008PTGastrinoma malignant10051709PTGastroenteropancreatic neuroendocrine tumour disease10077559PTGastrointestinal adenocarcinoma10081003PTGastrointestinal cancer metastatic10053548PT |
| Gastroenteropancreatic neuroendocrine tumour disease 10077559 PT Gastrointestinal adenocarcinoma 10081003 PT Gastrointestinal cancer metastatic 10053548 PT |
| Gastroenteropancreatic neuroendocrine tumour disease10077559PTGastrointestinal adenocarcinoma10081003PTGastrointestinal cancer metastatic10053548PT |
| Gastrointestinal cancer metastatic 10053548 PT |
| Gastrointestinal carcinoma 10017940 PT |
| Gastronitestinal caremonia |
| Gastrointestinal carcinoma in situ 10061168 PT |
| Gastrointestinal melanoma 10077167 PT |
| Gastrointestinal stromal cancer 10071653 PT |
| Gastrooesophageal cancer 10062878 PT |
| Genital cancer male 10073116 PT |
| Genital cancer male in situ 10073124 PT |
| Genital neoplasm malignant female 10018160 PT |
| Genitourinary melanoma 10077166 PT |
| Germ cell cancer 10061184 PT |
| Germ cell cancer metastatic 10068971 PT |
| Gestational trophoblastic tumour 10061988 PT |
| Gingival cancer 10067807 PT |


| NameCodeLevelMetastases to adrenals10027451PTMetastases to biliary tract10062195PTMetastases to bladder10049722PTMetastases to bone10027452PTMetastases to breast10027454PTMetastases to central nervous system10059282PTMetastases to chest wall10051663PTMetastases to diaphragm10051665PTMetastases to Eustachian tube10051666PT |
|---|
| Metastases to biliary tract10062195PTMetastases to bladder10049722PTMetastases to bone10027452PTMetastases to breast10027454PTMetastases to central nervous system10059282PTMetastases to chest wall10051663PTMetastases to diaphragm10051665PT |
| Metastases to bladder10049722PTMetastases to bone10027452PTMetastases to breast10027454PTMetastases to central nervous system10059282PTMetastases to chest wall10051663PTMetastases to diaphragm10051665PT |
| Metastases to bone10027452PTMetastases to breast10027454PTMetastases to central nervous system10059282PTMetastases to chest wall10051663PTMetastases to diaphragm10051665PT |
| Metastases to breast10027454PTMetastases to central nervous system10059282PTMetastases to chest wall10051663PTMetastases to diaphragm10051665PT |
| Metastases to central nervous system10059282PTMetastases to chest wall10051663PTMetastases to diaphragm10051665PT |
| Metastases to chest wall Metastases to diaphragm 10051663 PT 10051665 PT |
| Metastases to diaphragm 10051665 PT |
| Metastases to Eustachian tube 10051666 PT |
| Metastases to eye 10049724 PT |
| Metastases to fallopian tube 10049727 PT |
| Metastases to gallbladder 10051667 PT |
| Metastases to gastrointestinal tract 10062196 PT |
| Metastases to heart 10049717 PT |
| Metastases to kidney 10027455 PT |
| Metastases to larynx 10051668 PT |
| Metastases to liver 10027457 PT |
| Metastases to lung 10027458 PT |
| Metastases to meninges 10051696 PT |
| Metastases to mouth 10051669 PT |
| Metastases to muscle 10049730 PT |
| Metastases to nasal sinuses 10051670 PT |
| Metastases to neck 10027460 PT |
| Metastases to nervous system 10061287 PT |
| Metastases to oesophagus 10051671 PT |
| Metastases to ovary 10027462 PT |
| Metastases to pancreas 10049721 PT |
| Metastases to pelvis 10070913 PT |
| Metastases to penis 10051672 PT |
| Metastases to perineum 10051673 PT |
| Metastases to peripheral nervous system 10051674 PT |
| Metastases to peripheral vascular system 10058307 PT |
| Metastases to peritoneum 10051676 PT |
| Metastases to pharynx 10051677 PT |
| Metastases to pituitary gland 10049728 PT |
| Metastases to placenta 10049725 PT |
| Metastases to pleura 10027463 PT |
| Metastases to prostate 10051678 PT |
| Metastases to rectum 10051679 PT |
| Metastases to reproductive organ 10061288 PT |
| Metastases to retroperitoneum 10051680 PT |
| Metastases to salivary gland 10051681 PT |
| Metastases to skin 10027465 PT |
| Metastases to soft tissue 10062197 PT |


| NameCodeLevelPseudosarcoma10051807PT |
|-------------------------------------------------|
| 1364634160114 |
| Queyrat erythroplasia 10037732 PT |
| Rectal adenocarcinoma 10038019 PT |
| Rectal cancer 10038038 PT |
| Rectal cancer metastatic 10055097 PT |
| Rectal cancer recurrent 10038046 PT |
| Rectal cancer stage 0 10038047 PT |
| Rectal cancer stage I 10038048 PT |
| Rectal cancer stage II 10038049 PT |
| Rectal cancer stage III 10038050 PT |
| Rectal cancer stage IV 10038051 PT |
| Rectosigmoid cancer 10038086 PT |
| Rectosigmoid cancer metastatic 10069728 PT |
| Rectosigmoid cancer recurrent 10038094 PT |
| Rectosigmoid cancer stage 0 10038095 PT |
| Rectosigmoid cancer stage I 10038096 PT |
| Rectosigmoid cancer stage II 10038097 PT |
| Rectosigmoid cancer stage III 10038098 PT |
| Rectosigmoid cancer stage IV 10038099 PT |
| Recurrent cancer 10038111 PT |
| Refractory cancer 10070308 PT |
| Renal cancer 10038389 PT |
| Renal cancer metastatic 10050018 PT |
| Renal cancer recurrent 10038390 PT |
| Renal cancer stage I 10038391 PT |
| Renal cancer stage II 10038392 PT |
| Renal cancer stage III 10038393 PT |
| Renal cancer stage IV 10038394 PT |
| Renal cell carcinoma 10067946 PT |
| Renal cell carcinoma recurrent 10038410 PT |
| Renal cell carcinoma stage I 10038411 PT |
| Renal cell carcinoma stage II 10038412 PT |
| Renal cell carcinoma stage III 10038413 PT |
| Renal cell carcinoma stage IV 10038414 PT |
| Respiratory tract carcinoma in situ 10038724 PT |
| Retinal melanoma 10038878 PT |
| Retinoblastoma 10038916 PT |
| Retroperitoneal cancer 10038977 PT |
| Retroperitoneal neoplasm metastatic 10062485 PT |
| Rhabdoid tumour 10073334 PT |
| Rhabdoid tumour of the kidney 10039019 PT |
| Rhabdomyosarcoma 10039022 PT |
| Rhabdomyosarcoma recurrent 10039027 PT |
| Round cell liposarcoma 10073139 PT |


# 18.6 AESI: Malignancies

Events pertaining to PTs from MedDRA SMQ "Malignant or unspecified tumors" with rationales for inclusion/exclusion in the AESIs Malignancies.

| Origin<br>al<br>Study<br>Identifi<br>er | Subject<br>Identifie<br>r<br>(SUBJID | Unique Subject<br>Identifier<br>(USUBJID) | Study<br>Identifier<br>for AE<br>Occurence<br>(\$TUDYID) | Reported Term<br>(AETERM) | Dictionary-<br>Derived<br>Term<br>(AEDECOD) | Start Date/Tim e of Adverse Event (AESTDT C) | End Date/Tim e of Adverse Event (AEENDT C) | Severity/<br>Intensity<br>(AESEV) | Reported<br>Causalit<br>y<br>(AEREL) | Outcome of Adverse<br>Event (AEOUT) | SMQ<br>Malignan<br>t or<br>unspecifi<br>ed<br>tumors | AESI =<br>Maligna<br>nt<br>tumors | Rationale for exclusion | Data<br>Sour<br>ce |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| PPD | | | | | | | | | | | | | | |













# **ELECTRONIC SIGNATURES**

# Document: emr 700568-012-integrated analysis plan-text-final-v 1

| Signed By Event Name | | Meaning of Signature | Server Date<br>(dd-MMM-yyyy<br>HH:mm 'GMT'Z) |
|---|---|---|---|
| PPD | Task Completed (Approval eSign): Approved | Business Approval | 11/22/2018 02:15:01 |